

Protocol version: 9



Transcranial Direct Current Stimulation in Major Depressive Disorder: a Double-blind, Placebo-controlled, Randomized, Superiority Trial

**Protocol Number: FL001** 

Version: 9

**Date: 10Jan2023** 

Sponsor:

Flow Neuroscience AB

Södra Förstadsgatan 2, 211 43 Malmö

Phone: +46736607170

**Sponsor Contact:** 

Erik Rehn

Chief Technology Officer & Co-Founder

Email: erik@flowneuroscience.com

Phone: +46736607170

This document contains confidential information for use only by investigators participating in the clinical investigation. This document should be maintained in a secure location and should not be copied or made available for review by unauthorized personnel.

Protocol version: 9



# 2 REVISION HISTORY

| Version | Date | Summary of Changes |
|---|---|---|
| 1.0 | 10 Nov 2021 | First Version for IDE submission |
| 2 | 26 Nov 2021 | <ul> <li>Removed upper age limit.</li> <li>MADRS-s of 20 or above added to inclusion criteria.</li> <li>Improved references.</li> <li>Clarified that the participants must be living in England, Wales or Texas.</li> <li>Added optional early termination visit.</li> </ul> |
| 2 | 13 Dec 2021 | Incorporation of FDA comments from IDE application SDMT baseline moved to week 0 visit. |
| 2 | 05 Jan 2022 | - Change to PHQ-9 form MADRS-s for the first screening assessment after consent PHQ-9 of 10 points or above added to inclusion criteria MADRS-s of 20 or above removed from inclusion criteria. |
| 3 | 19Feb2022 | <ul> <li>Inclusion criteria 12 update age to ≥ age 18</li> <li>Exclusion criteria 28 updated to: Are a chronic tobacco smoker, as defined by smoking by smoking &gt;100 cigarettes (including hand-rolled cigarettes, cigars, cigarillos, etc.) in their life-time and have smoked every day for the last 7 days.</li> </ul> |
| 4 | 23Feb2022 | <ul> <li>Updated exclusion criteria 31 to: Are participating concurrently in another clinical investigation or have participated in a clinical investigation within the last 90 days or intend to Participate in another clinical investigation during the study, and where the participation in the other investigation might interfere with the results of this trial as deemed by the PI.</li> <li>Clarified that for inclusion criteria 11 the age is 18 for UK and 22 for the US.</li> </ul> |
| 5 | 16Mar2022 | - Updated device traceability (section 8.3) to reflect that UK participants are allowed to keep the device after trial completion. |
| 6 | 04Apr2022 | - Removed PHQ-9 from screening Clarified which AEs will be followed-up in more detail. Anticipated AEs will be recorded using AEQ Moved some sections regarding how missing data is handled in the statistical analysis plan to a new document (Statistical analysis plan - FL001) Site staff will consent subjects not Curebase staff. |





| 7 | 31Aug2022 | <ul> <li>Clarified insomnia &amp; sleep apnea as an exclusion criteria, added eating disorders.</li> <li>Changed some excl. criteria based comorbidities to not be life-long.</li> <li>Clarified primary endpoint as requested by FDA IDE feedback.</li> </ul> |
|---|---|---|
| 8 | 07Dec2022 | <ul> <li>Added reference to adaptive design report (22.15)</li> <li>Updated primary endpoint formulation again as requested by the FDA.</li> <li>EQ-5D-3L is now a secondary endpoint as requested by the FDA.</li> <li>Added within-patient clinically meaningful change exploratory endpoint.</li> <li>Added clarification of when the randomization happens (22.4)</li> <li>Added section 13.4 describing routines regarding video calls, as requested by the FDA.</li> </ul> |
| 9 | 10Jan2023 | <ul> <li>Removed need for CRO representative to sign this<br/>protocol since they are not involved in the development<br/>of this protocol.</li> </ul> |



Protocol version: 9



## 3 PROTOCOL APPROVAL SIGNATURE PAGE

Protocol Number: FL001 Protocol Version: 9 Protocol Date: 10Jan2023

Protocol Name: Transcranial Direct Current Stimulation in Major Depressive Disorder: A

Double-blind, Placebo-controlled, Randomized, Superiority Trial

This protocol has been read and approved by:

| SPONSOR: | |
|---|---|
| Erik Rehn<br>Chief Technology Officer & Co-Founder<br>Flow Neuroscience AB | Signature & Date: |



Protocol version: 9



#### 4 INVESTIGATOR PROTOCOL SIGNATURE PAGE

The signature below documents the receipt and review of the Study Protocol and any attachments and provides the necessary assurances that this study will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to the local legal and regulatory requirements and applicable United States Federal Regulations, ISO 14155:2020, ICH and GCP guidelines, and the latest version of the Declaration of Helsinki.

I have read and understand this protocol and will conduct the study in accordance with this protocol, all attachments and amendments, applicable Food and Drug Administration regulations, HIPAA, IRB/EC requirements, and the policies of the institutions where the study will take place.

In my formal capacity as Investigator, my duties include ensuring the safety of the study subjects enrolled under my supervision and providing Flow Neuroscience AB with complete and timely information, as outlined in the protocol. It is understood that all information pertaining to the study will be held strictly

| Protocol Number: FL001 | Protocol Version: 9 | Protocol Date: 10jan2023 |
|---|---|---|
| Protocol Name: Transcranial Dire Placebo-controlled, Randomized, | | or Depressive Disorder: A Double-blind, |
| Investigator: | | |
| (Print Name) | | |
| (Signature) | | Date (dd/mmm/yyyy) |
| Sponsor Representative Name | | |
| Sponsor Signature | | Date (dd/mmm/yyyy) |
| Legal Representative Name | | |
| Legal Representative Signature | | Date (dd/mmm/yyyy) |
| Upon signing, send a copy of this | page to Curebase and retain | a copy for your files. |





# TABLE OF CONTENTS

| 1 TITLE PAGE | 1 |
|---|---|
| 2 REVISION HISTORY | 2 |
| 3 PROTOCOL APPROVAL SIGNATURE PAGE | 4 |
| 4 INVESTIGATOR PROTOCOL SIGNATURE PAGE | 5 |
| 5 LIST OF ABBREVIATIONS | 10 |
| 6 Study Summary | 12 |
| 7 Schedule of Procedures | 19 |
| 8.1 Background 8.1.1 Major Depressive Disorder (MDD) 8.1.2 MDD Diagnosis 8.1.3 Other Treatment Options 8.1.3.1 Antidepressants 8.1.3.2 Psychological Treatments 8.1.3.3 Electroconvulsive Therapy (ECT) 8.1.3.4 Transcranial Magnetic Stimulation (TMS) 8.1.3.5 Cranial Electrotherapy Stimulation (CES) 8.1.3.6 Transcranial Direct Current Stimulation (tDCS) 8.2 Investigational Device 8.2.1 Flow FL-100 8.2.2 The Flow app 8.3 Device Traceability 8.4 Supply and Accountability of Investigational Devices 8.5 Device Use Experience and Training | 21 21 21 21 21 21 21 23 23 24 24 24 25 25 26 28 29 |
| 9 Benefit-Risk Analysis 9.1 Risks 9.2 Risk Mitigation 9.2.1 Monitors 9.2.2 Stimulation Parameter Space 9.2.3 Usage Limits 9.3 Anticipated Benefits 9.4 Risk-to-Benefit Ratio | 29<br>29<br>30<br>31<br>31<br>31<br>31 |
| 10 Study Objectives 10.1 Background | <b>31</b><br>31 |





| 12.5 Screen Failures | 38 |
|-----------------------------------------------------------|----------|
| 12.4.1 Participant Enrollment 12.5 Screen Failures | 38<br>38 |
| · | |
| · | |
| 12.6 Participant Treatment Assignment | 39 |
| 12.0 Participant Treatment Assignment | 39 |
| 13 Study Procedures | 39 |
| 13.1 Week -3 to -1: Informed Consent (ICF) | 39 |
| 13.2 Week 0 | 40 |
| 13.3 Weeks 1, 4 & 7 | 40 |
| 13.4 Week 10 | 41 |
| 13.5 Week 20 Follow-Up Visit - Open-Label Only | 41 |
| 13.6 Video calls | 42 |
| 13.7 Late and Missed Visits | 42 |
| 13.8 Unscheduled Visits | 43 |
| 13.9 Study Completion/Discontinuation | 43 |
| 10.9 Study Completion/Discontinuation | 43 |
| 14 Description of Study Procedures | 43 |
| 15 Early Discontinuation: Participants | 45 |
| 15.1 Technical Failures | 45 |
| 15.2 Treatment Failures | 45 |
| 15.3 Lost to Follow-Up (LTFU) | 46 |
| • • • • | |
| 15.4 Withdrawals | 46 |
| 15.5 Documentation of Early Discontinuation and Pregnancy | 47 |
| 15.6 Use of Data from Early Discontinuation Cases | 47 |
| 15.7 Ongoing Treatment for Early Discontinuation Cases | 47 |
| 16 Early Discontinuation: Study | 47 |





| 16.3 Routine Close-Out 17 Protocol Deviations 18 Concomitant Medications/Therapies 19 Adverse Event & Device Deficiency Reporting 19.1 Definitions 19.2 Classification of an AE 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.3 Itudy Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | 16.1 Procedure for Suspension or Early Termination | 47 |
|---|---|---|---|
| 18 Concomitant Medications/Therapies 19 Adverse Event & Device Deficiency Reporting 19.1 Definitions 19.2 Classification of an AE 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (ITT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5 Tovariates/Covariate Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 48<br>48 |
| 18 Concomitant Medications/Therapies 19 Adverse Event & Device Deficiency Reporting 19.1 Definitions 19.2 Classification of an AE 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (ITT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5 Tovariates/Covariate Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | |
| 19 Adverse Event & Device Deficiency Reporting 19.1 Definitions 19.2 Classification of an AE 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5 Tovariates/Covariate Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | 17 | Protocol Deviations | 48 |
| 19.1 Definitions 19.2 Classification of an AE 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | 18 | Concomitant Medications/Therapies | 49 |
| 19.2 Classification of an AE 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis | 19 | | 49 |
| 19.2.1 Severity 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis | | | 50 |
| 19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3.3 flutent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5 Missing Data/Sensitivity Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis | | | 52 |
| 19.2.3 SAE Relationship Assessment 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis | | • | 52 |
| 19.2.4 SAE Reporting 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 AS Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis | | · | 52 |
| 19.2.5 Determination and Reporting of Unanticipated Adverse Device Effects (US Sites) 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5 Missing Data/Sensitivity Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis | | · | 52 |
| 19.3 Treatment of AEs 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 54 |
| 19.4 Safety Oversight: Clinical Events Committee (CEC) 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | · | 55 |
| 19.5 Safety/Suicide Risk Management Plan 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 55 |
| 20 Stopping rules 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 55 |
| 21 Clinical Monitoring 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | 19.5 Safety/Suicide Risk Management Plan | 55 |
| 21.1 Site Monitoring 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | 20 | Stopping rules | 56 |
| 21.2 Monitoring Activities 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | 21 | Clinical Monitoring | 56 |
| 21.3 Frequency of Visits 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | 21.1 Site Monitoring | 56 |
| 21.4 Audit and Inspections 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | 21.2 Monitoring Activities | 57 |
| 22 Statistical analysis 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | 21.3 Frequency of Visits | 58 |
| 22.1 Study Hypothesis 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | 21.4 Audit and Inspections | 58 |
| 22.2 Sample Size Assumptions and Calculations 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | 22 | Statistical analysis | 59 |
| 22.3 Study Populations 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | • • • | 59 |
| 22.3.1 Intent-to-Treat Analysis Set (ITT) 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | · | 59 |
| 22.3.2 As Treated Analysis Set (AT) 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | · | 59 |
| 22.3.3 Modified Intent-to-Treat Analysis Set (mITT) 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | • , , | 59 |
| 22.3.4 Per Protocol Analysis Set (PP) 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 59 |
| 22.4 Randomization 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | · | 59 |
| 22.5 Testing of Primary Effectiveness Hypotheses 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | · | 60 |
| 22.5.1 Multiple Imputation Analysis 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 60 |
| 22.6 Missing Data/Sensitivity Analysis 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 60 |
| 22.7 Covariates/Covariate Analysis 22.8 Secondary Effectiveness Endpoints | | | 61 |
| 22.8 Secondary Effectiveness Endpoints | | | 61<br>61 |
| · | | · | 61<br>61 |
| 22.9 Exploratory Engloritis | | | 61<br>62 |
| | | 22.9 Exploratory Enupolitis | 62 |



# Clinical Study Protocol

T1 Effective Date: 19FEB2021

| 22.10 Multiplicity Adjustment | 62 |
|-------------------------------------------|----|
| 22.11 Evaluation of Blinding | 63 |
| 22.12 Device Survival | 63 |
| 22.13 Poolability Analysis | 63 |
| 22.14 Safety Analyses | 63 |
| 22.15 Interim Analyses | 64 |
| 23 Ethics & Protection of Human Subjects | 64 |
| 23.1 Ethical Review | 64 |
| 23.2 Regulatory Considerations | 64 |
| 23.3 Study Amendments | 65 |
| 23.4 Insurance | 65 |
| 24 Data Handling and Recordkeeping | 65 |
| 24.1 EDC and eCRFs | 65 |
| 24.2 Capture of patient reported outcomes | 66 |
| 24.3 Study Records Retention | 66 |
| 24.4 Publication and Data Sharing Policy | 67 |
| 24.5 Participant and Data Confidentiality | 67 |
| 24.6 Investigator Records | 68 |
| 24.7 Participant Records | 68 |
| 24.8 Investigator Records and Reports | 68 |



Protocol version: 9



### 5 LIST OF ABBREVIATIONS

ADE Adverse Device Effect

**AE** Adverse Event

AEQ tDCS Adverse Events Questionnaire
ATHF Antidepressant Treatment History Form
ATT Average Treatment effect on the Treated

**CA** Competent Authority

**CABG** Coronary Artery Bypass Graft

**CDC** Center for Disease Control and Prevention

**CEC** Clinical Events Committee

CFR Code of Federal Regulations
CHF Coronary Heart Failure

CMP Clinical Monitoring Plan

CRO Contract Research Organization
ClinRO Clinician Reported Outcome

**C-SSRS** Columbia Suicide Severity Rating Scale

**DBS** Deep Brain Stimulation

**DHHS**U.S. Department of Health and Human Services

**DLPFC** Dorsolateral Prefrontal Cortex

**DMP** Data Management Plan

**EC** Ethics Committee

eCRF Electronic Case Report Form
ECT Electroconvulsive Therapy
EDC Electronic Data Capture
EOB Explanation of Benefits

**FDA** U.S. Food and Drug Administration

GCP Good Clinical Practice

HAM-A Hamilton Anxiety Rating ScaleHDRS-17 Hamilton Depression Rating Score

HIPAA Health Insurance Portability and Accountability Act

ICF Informed Consent Form

International Conference on Harmonization of Technical Requirements

for Registration of Pharmaceuticals for Human Use

IDE Investigational Device Exemption

**IFU** Instructions for Use

iOS iPhone Operating SystemIRB Institutional Review BoardISF Investigator Site File



Protocol version: 9



ITT Intent-to-Treat
LB Lower Bound
LTFU Lost to Follow-Up

MADRS Montgomery–Åsberg Depression Rating Scale

MADRS-s Montgomery—Asberg Depression Rating Scale - Self-report

MAOIs Monoamine oxidase inhibitors
MDD Major Depressive Disorder

MI Multiple Imputation

MINI Mini International Neuropsychiatric Interview

NASSA Noradrenaline and Specific Serotonergic Antidepressant

mITT Modified Intent to Treat
NRS Numeric Rating Scale

NSAIDS Nonsteroidal anti-inflammatory drugs
OCD Obsessive-Compulsive Disorder

OHRP U.S. Office of Human Research Protections

PMA Premarket Approval

**PP** Per-Protocol

PRO Patient Reported Outcome

PS Propensity Score
QOL Quality of Life

**RAVLT** Rey Auditory Verbal Learning Test

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SDMT Symbol-Digit Modalities Test
SDW Source Document Worksheet
SMD Standardized Mean Differences

**SNRI** Serotonin and Noradrenaline Reuptake Inhibitor

**SOC** Standard of Care

**SSRI** Selective Serotonin Reuptake Inhibitor

**SOP** Standard Operating Procedure

**TAQ** Treatment Acceptability Questionnaire

TCA Tricyclic Antidepressant

Transcranial Direct Current Stimulation
TEM Treatment-Emergent Mania/hypomania
TMS Transcranial Magnetic Stimulation
UADE Unanticipated Adverse Device Effect

**UB** Upper Bound

WHO World Health Organization
YMRS Young Mania Rating Scale

Protocol version: 9



# 6 STUDY SUMMARY

| Study Full Title | Transcranial Direct Current Stimulation in Major Depressive Disorder: A Double-blind, Placebo-controlled, Randomized, Superiority Trial |
|---|---|
| Study Sponsor | Flow Neuroscience AB |
| Study Number | FL001 |
| Device Name | Flow FL-100 |
| Protocol Date | 10Jan2023 |
| STUDY OVERVIEW | |
| Study Design | Double-blind, placebo-controlled, randomized, superiority, remote. |
| Purpose | The purpose of this trial is to investigate the use of the Flow FL-100 device at-home to treat Unipolar Major Depressive Disorder (MDD) in a double-blind RCT. |
| Expected Study Duration | 10 months |
| Evaluation Schedule | Participants will undergo evaluations at the following study visits. Various evaluations regarding depression severity, suicidal ideation will be performed (see Schedule of Evaluations for more detail): • Pre-Treatment Phase - Week -3 - Week -2 - Week -1 • Blinded Phase - Week 0 - Week 1 - Week 4 - Week 7 - Week 10 • Open-Label Phase - Week 20 At week 0, 1, 4, 7, 10, 20, participants will also complete the MADRS-s on their personal smartphone or other device running Android 5.0+ or iPhone Operating System (iOS) 12+. |
| ELIGIBILITY CRITERIA | |





| Intended Participant Population | Up to 270 participants will be randomized at 2 sites, one located in the United Kingdom and the other in the United States. The recruitment will be capped to 155 for each of the sites. |
|---|---|
| | 1:1 randomization: Flow FL-100 vs. Sham |
| | To be eligible to participate in this study, participants must meet all the following criteria: |
| | 1. Be ≥18 years. |
| | Have a diagnosis of Unipolar MDD with a current depressive episode as defined by the diagnostic criteria in the Diagnostic and statistical manual of mental disorders – 5th edition (DSM-V) |
| | <ol> <li>Have a Hamilton Depression Rating Score (HDRS-17) of ≥ 16.</li> </ol> |
| Diagnosis and Inclusion | 4. For 6 weeks prior to enrollment, are either: a. not taking antidepressant medication or: b. are taking a stable antidepressant regimen with a stable medication source and agree to continue the same regimen throughout study participation. 5. If in psychotherapy, have maintained stable |
| Criteria | psychotherapy for at least 6 weeks prior to enrollment. 6. Have access to a stable internet connection through |
| | which the treatment will be received. |
| | 7. Have access to a smartphone or other device running Android 5.0+ or iPhone Operating System (iOS) 12+ (e.g., reasonably new iPhone/iPad or Android phone), used to using the device in their everyday life, and can capably use the study application on the device, as determined by the investigator. |
| | 8. Are currently living in England/Wales (UK) or Texas (US). |
| | 9. Subject is currently under the care of a psychiatrist or a primary care physician, agrees to be evaluated at regular intervals by a psychiatrist or primary care physician for the duration of study participation, and agrees to promptly inform the study staff of any change of psychiatric or mental health providers during study participation. |





| | T |
|---|---|
| | <ul> <li>10. Subject agrees to allow any and all forms of communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within at least two years of study enrollment.</li> <li>11. Subject agrees to provide the name and verifiable contact information (email and mailing addresses, mobile and land-line phone numbers, as applicable) of at least two persons ≥ age 18 (22 in the US) who reside within a 60-minute drive of the patient's residence and whom the research staff is at liberty to contact, as they deem necessary, for the duration of study participation.</li> <li>12. Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study.</li> <li>13. Be willing and able to comply with all study procedures.</li> </ul> |
| | 14. Subject agrees to meet all of the inclusion criteria throughout their participation in the study. Otherwise, |
| | the subject will be discontinued from the study. 15. Subject agrees to a Safety/Suicide Risk Management Protocol, which is intended to reduce the reduce the risk of suicide during study participation. |
| | Participants who meet any of the following criteria will be excluded from participating in this study: |
| | <ol> <li>Are in a current state of mania, as determined by the YMRS or psychosis, as determined by the MINI.</li> <li>Are diagnosed with vitamin or hormonal deficiencies that may mimic mood disorders, as determined by the investigator.</li> </ol> |
| Exclusion Criteria | 3. Are currently receiving any other interventional therapy for MDD other than a stable regimen of antidepressants or psychotherapy as defined in the inclusion criteria. |
| | 4. Considered to have treatment resistant depression as defined by inadequate clinical response to 2 or more trials of antidepressants at an adequate dose and duration. |
| | Have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), cranial |





- electrotherapy stimulation (CES), transcranial direct current stimulation (tDCS), deep brain stimulation (DBS), or other brain stimulation.
- 6. Patient answers Yes to Questions 4, 5 or 6 on the Columbia Suicide Severity Rating Scale (C-SSRS) Triage and Risk Identification Screener.
- 7. Any previous hospitilization for suicidal behavior.
- 8. Have chronic severe insomnia (< 4 hours of sleep each night), or depression secondary to chronic insomnia or sleep apnea.
- 9. Have any structural lesion (e.g., any structural neurological condition, or more subcortical lesions than would be expected for age or have had a stroke that affects stimulated area or connected areas) or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results, as determined by the investigator.
- Have any implant in the brain (e.g., DBS) or neurocranium, or any other active implantable medical device.
- 11. Have any neurocranial defect.
- 12. Have a history of epilepsy or seizures (including history of withdrawal / provoked seizures).
- 13. Have shrapnel or any ferromagnetic material in the head.
- 14. Have any disorder that would impair the ability to complete the study questionnaires.
- 15. Have been diagnosed with autism spectrum disorder.
- 16. Are actively abusing substances (<1 week prior to enrollment).
- 17. Have a cognitive impairment (including dementia).
- 18. Have a history of mania or psychosis.
- 19. Are currently using any medications that affect cortical excitability (e.g., benzodiazepines, epileptics, etc.).
- 20. Are currently experiencing symptoms of withdrawal from alcohol or benzodiazepines.
- 21. Have been diagnosed with Parkinsonism or other movement disorder as determined by the investigator to interfere with treatment.





- 22. Have ever taken esketamine / ketamine for treatment of depression.
- 23. Have ever been admitted to hospital for depression.
- 24. Have ever been diagnosed with obsessive-compulsive disorder (OCD) or bipolar type 1 or 2 disorder.
- 25. Is diagnosed with an active primary anxiety disorder, or PTSD, agoraphobia, anorexia or bulimia, panic or personality disorder with active symptoms.
- 26. Have a history of psychosurgery for depression.
- 27. Have any history of myocardial infarction, coronary artery bypass graft (CABG), coronary heart failure (CHF), or history of other cardiac issues.
- 28. Are currently experiencing or have a history of intractable migraines.
- 29. Are a chronic tobacco smoker, as defined by smoking by smoking >100 cigarettes (including hand-rolled cigarettes, cigars, cigarillos, etc.) in their life-time and have smoked every day for the last 7 days.
- 30. If female and of child-bearing potential, currently pregnant or breastfeeding or planning to become pregnant or breastfeed any time during the study.
- 31. Are currently a prisoner.
- 32. Are participating concurrently in another clinical investigation or have participated in a clinical investigation within the last 90 days or intend to Participate in another clinical investigation during the study, and where the participation in the other investigation might interfere with the results of this trial as deemed by the PI.
- 33. Have any medical condition or other circumstances, in the judgment of the investigator, that might interfere with the ability to complete follow-up visits and the self-reported MADRS-s in the app.
- 34. Have any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the device's safety and performance.
- 35. A Subject who meets any of the exclusion criteria during study participation will be discontinued from the study.





| FL-100 treatment sessions | FL-100 will be used by patients remotely for five sessions per week for 3 weeks, followed by three sessions per week for 7 weeks. In total, thirty-six sessions over 10 weeks during the blinded phase. |
|---|---|
| STUDY ENDPOINTS | |
| Primary Endpoint | The primary effectiveness endpoint is the adjusted mean group difference in the HDRS-17 scores at 10 weeks compared to baseline for subjects in the Active device and the Sham device groups. |
| Secondary Endpoints | <ul> <li>Arm difference in HDRS-17 response and remission rate at week 10.</li> <li>Arm difference in MADRS average score change, and response and remission rate at week 10.</li> <li>Arm difference in MADRS-s average score change, and response and remission rate at week 10.</li> <li>Quality of life improvement as measured by EQ-5D-3L in the active compared to sham arm at week 10.</li> </ul> |
| Exploratory Endpoints | <ul> <li>Young Mania Rating Scale (YMRS) at 10 weeks.</li> <li>tDCS Adverse Events Questionnaire (AEQ) at 10 and 20 weeks</li> <li>Hamilton Anxiety Rating Scale (HAM-A) change at week 10.</li> <li>HDRS-17, MADRS, MADRS-s mean decrease, and remission and response rate at 20 weeks (after open-label) compared to open-label start and baseline.</li> <li>Correlation between MADRS and MADRS-s.</li> <li>Correlation between adherence to stimulation and HDRS-17/MADRS decrease in the active group at 10 weeks.</li> <li>Neuropsychological measure: verbal learning (Rey Auditory Verbal Learning Test (RAVLT) and information processing speed (Symbol-Digit Modalities Test (SDMT)</li> <li>Treatment acceptability questionnaire (TAQ) as developed by UEL. There is one form at baseline and another at week 10 and 20.</li> <li>The within-patient clinically meaningful improvement as defined as at least -3 points on the HDRS-17 scale. The percentage of subjects for each arm that</li> </ul> |





| | reaches -3 points or more improvement and also the Cumulative Distribution Function Curves of Change in HDRS-17 Score from Baseline to Primary end-point by arm. |
|---|---|
| STATISTICAL CONSIDERATION | |
| Sample Size | 270 |
| Statistical Plan | A modified intent to treat will be used. Users who have performed less than 10 sessions (300 minutes) during the first 3 weeks will be excluded from the analysis. |
| STUDY MANAGEMENT | |
| Principal Investigator UK | Professor of Affective Neuroscience Cynthia Fu, MD, PhD, University East London |
| Principal Investigator US | Associate Professor of Psychiatry Sudhakar Selvaraj, MD, PhD, University of Texas |
| Clinical Research Organization (CRO) | Curebase, Inc. |

Protocol version: 9



# 7 Schedule of Procedures

Table 1. Schedule of Procedures. Activities in blue cells are performed by trained graduate researchers supervised by a trained psychiatrist, and red cells are to be completed by the participant.

| | Pre-Treatme<br>nt | | E | Blinded Pha | Open-Label<br>Phase | | Early termination <sup>8</sup> | | |
|---|---|---|---|---|---|---|---|---|---|
| Activity | Week<br>-3 to -1<br>(± 3 days) | Week<br>0 | Week 1<br>(± 3<br>days) | Week 4<br>(± 3<br>days) | Week<br>7<br>(± 3<br>days) | Week 10<br>(± 3 days)<br>Final<br>blinded<br>visit <sup>1</sup> | Week 10<br>(± 3<br>days)<br>Open<br>Label<br>Start | Wee<br>k 20<br>(± 3<br>days) | Week 1-20 |
| Informed<br>Consent | X | | | | | | | | |
| Screening and baseline Video Call | Х | | | | | | | | |
| Diagnostic<br>Assessment for<br>MDD | Xa | | | | | | | | |
| Intervention Kit<br>Shipped to<br>subject | X <sup>5</sup> | | | | | | | | |
| Randomization <sup>6</sup> | | Х | | | | | | | |
| Technical onboarding | | Х | | | | | | | |
| Initial Visit | | Χ | | | | | | | |
| Video call | Х | Х | Х | Х | Х | Х | | Х | Х |
| MINI | Х | | | | | | | | |
| HDRS-17 | X | | Х | Х | Х | Х | | Х | X |
| MADRS | Х | > 11 | X | X | X | X | | X | X |
| MADRS-s | V | X <sup>4</sup> | X | X | X | X | | X | X |
| C-SSRS | X | | X | X | X | X | | X | X |
| YMRS | X | | Х | Х | Х | X | | X | X |
| HAM-A | X | | | | | X | | X | X |
| EQ-5D-3L<br>RAVLT | X | | | | | X | | X | X |
| SDMT | X | X <sup>2</sup> | | | | X X <sup>2</sup> | | X<br>X <sup>2</sup> | ۸ |
| TAQ | X | ^ | | | | X | | X | Х |
| AEQ | A | | | | | X | | X | X |
| Healthcare Visit | | | | | | | | | |
| Survey <sup>3</sup> | | | | | | Х | | X | X |
| FLOW FL-100 use <sup>7</sup> | | Х | Х | Х | Х | Х | Х | Х | |
| Record/Review<br>Concomitant<br>Medications | Х | Х | Х | Х | Х | х | | Х | х |
| Record/Review<br>Adverse Events | | Х | Х | Х | Х | Х | | Х | Х |



Protocol version: 9



<sup>1</sup> The week 10 visit includes the study Primary end-point. This will be the final blinded visit and will be the start of the open label phase of the study. Participants in the Sham arm will be informed of their assignment and will restart with active stimulation for 10 weeks; participants in the Flow FL-100 arm will be allowed to continue maintenance treatment for 10 more weeks at 3 sessions per week. The unblinding will occur after the primary end-point data has been recorded.
<sup>2</sup> Optional

Table 2. Stimulation schedule during blinded phase.

| Week | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|--------------------|---|---|---|---|---|---|---|---|---|----|
| Number of sessions | 5 | 5 | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |

Table 3. Stimulation schedule during open-label phase.

| Week | Previous<br>assignm<br>ent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of | Active | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |
| sessions | Sham | 5 | 5 | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |

<sup>&</sup>lt;sup>3</sup> Participants will be surveyed about the number of times he/she has sought healthcare due to depression during the previous 10 weeks.

<sup>&</sup>lt;sup>4</sup> Participants will be required to answer the nine questions of the MADRS-s form in the app to start the first stimulation session during the technical onboarding.

<sup>&</sup>lt;sup>5</sup> Participants will be required to start treatment within 24 days from completing the baseline surveys.

<sup>&</sup>lt;sup>6</sup> Completed after eligibility is confirmed by the investigator; when the participant signs up with their email in the trial app they will automatically be randomized to the sham or active treatment arm (with 50% probability).

<sup>&</sup>lt;sup>7</sup> Five sessions per week for 3 weeks, followed by three sessions per week for 7 weeks. In total, thirty-six sessions during 10 weeks during the blinded phase. Please refer to Table 2 and Table 3 below for more details.

<sup>&</sup>lt;sup>8</sup> In case there is an early termination the research staff can request to have an early termination interview, if the subject agrees.

<sup>9</sup> Diagnostic Assessment for MDD will be performed by Investigator-Psychiatrist according to the most recent APA Practice Guideline for treatment of MDD.

Protocol version: 9



# 8 Introduction

#### 8.1 BACKGROUND

#### 8.1.1 Major Depressive Disorder (MDD)

Major depressive disorder (MDD) is a common psychiatric condition, mostly treated with antidepressant drugs, which are limited for issues such as effectiveness and adverse effects.

#### 8.1.2 MDD DIAGNOSIS

The diagnosis of MDD is based on the diagnostic criteria in the Diagnostic and statistical manual of mental disorders – 5th edition (DSM-V). Patients should receive a thorough diagnostic assessment in order to establish the diagnosis of major depressive disorder, identify other psychiatric or general medical conditions that may require attention. The psychiatrist should develop a comprehensive plan for treatment. This evaluation generally includes a history of the present illness and current symptoms that may trigger or exacerbate depressive symptoms. Several clinically validated standard scales are available for the assessment of the severity of depressive symptoms. Based on cut-offs from these scales, the severity of MDD can be classified as mild, moderate, and severe.

#### 8.1.3 OTHER TREATMENT OPTIONS

#### 8.1.3.1 Antidepressants

Antidepressants are psychiatric drugs used for the treatment of MDD and other conditions, including dysthymia, anxiety disorders, OCD, eating disorders, chronic pain, neuropathic pain and, in some cases, dysmenorrhea, attention-deficit hyperactivity disorder, addiction, and sleep disorders. They may be prescribed alone or in combination with other medications. The Center for Disease Control and Prevention (CDC) reported that antidepressant usage in the United States among people aged 12 or more years rose by 400% between 1988-1994 and 2005-2008. Antidepressants are given to improve depressive symptoms.

There are several types of antidepressants, depending to the main neurotransmitter system they target:

Selective Serotonin Reuptake Inhibitors (SSRIs) and Serotonin and Noradrenaline
 Reuptake Inhibitors (SNRIs): SSRIs and SNRIs block the reuptake of serotonin or serotonin
 and noradrenaline in the brain. SSRIs are more widely prescribed than SNRIs, are effective
 in treating depression, and have fewer side-effects than older antidepressant classes <sup>1</sup>.
 One of the largest studies on MDD to date, the STAR\*D study, showed remission rates up

<sup>&</sup>lt;sup>1</sup> Anderson HD, Pace WD, Libby AM, West DR, Valuck RJ. Rates of 5 common antidepressant side effects among new adult and adolescent cases of depression: a retrospective US claims study. Clin Ther. 2012 Jan;34(1):113-23. doi: 10.1016/j.clinthera.2011.11.024.

Protocol version: 9



- to 28% with SSRIs alone <sup>2</sup>. SSRIs and SNRIs may have the following side effects: hypoglycemia, low sodium, nausea, rash, dry mouth, constipation, diarrhea, weight loss, sweating, tremor, sedation, sexual dysfunction, insomnia, headache, dizziness, anxiety, agitation, and abnormal thinking.
- Monoamine oxidase inhibitors (MAOIs): MAOIs inhibit the action of monoamine oxidase, the enzyme that breaks down monoaminergic neurotransmitter (e.g., serotonin, noradrenaline), thus increasing their levels in the brain. MAOIs are usually prescribed as second-line antidepressants as they present several side effects including blurred vision, rash, seizures, edema, weight disturbances, sexual dysfunction, diarrhea, nausea, constipation, anxiety, insomnia, drowsiness, headache, dizziness, arrhythmia, fainting and hypertension.
- <u>Noradrenaline and Specific Serotonergic Antidepressants (NASSAs)</u>: This class of antidepressants block adrenergic and specific serotonergic receptors. NASSAs have the following side effects: constipation, dry mouth, weight gain, drowsiness, sedation, blurred vision, and dizziness. More serious adverse reactions include seizures, white blood cell reduction, fainting, and allergic reactions.
- <u>Tricyclic Antidepressants (TCA):</u> This is the oldest class of antidepressants which are not typically used as first-line treatment because they have a less favorable tolerability and safety profile than more recent antidepressants. TCAsmay have the following side effects: seizures, insomnia, anxiety, arrhythmia, hypertension, rash, nausea, vomiting, abdominal cramps, weight loss, constipation, urinary retention, eye pressure, and sexual dysfunction.

Current practice for selecting pharmacological antidepressant treatments are limited by low response and remission rates in MDD. The UK National Institute for Health and Care Excellence (NICE) CG90 guidelines<sup>3</sup> indicate that antidepressants should not be routinely used for the initial treatment of mild depression, because the risk-benefit ratio is poor. Antidepressant treatment should be considered for people with a history of moderate or severe depression, and for those with mild depression that has been present for a long period.

The guidelines further note that antidepressant treatment should be used in combination with psychosocial interventions, should be continued for at least six months to reduce the risk of relapse, and that SSRIs are typically better tolerated than other antidepressants<sup>4</sup>. The American

<sup>&</sup>lt;sup>2</sup> Sinyor M, Schaffer A, Levitt A. The sequenced treatment alternatives to relieve depression (STAR\*D) trial: a review. Can J Psychiatry. 2010 Mar;55(3):126-35. doi: 10.1177/070674371005500303.

<sup>&</sup>lt;sup>3</sup> Depression: The treatment and Management of depression in adults (updated edition)" NICE guidelines [CG90].

<sup>&</sup>lt;sup>4</sup> Depression: The treatment and Management of depression in adults (updated edition)" NICE guidelines [CG90].

Protocol version: 9



Psychiatric Association treatment guidelines<sup>5</sup> recommend antidepressant medication as an initial treatment choice in people with mild or moderate major depression and should be given to all patients with severe depression. Moreover, treatment should be individually tailored and should consider all available options that may include pharmacotherapy (other symptomatic treatments), psychotherapy, ECT, TMS or tDCS.

# 8.1.3.2 Psychological Treatments

Many psychological treatments are available for MDD. These include but not limited to, psychoeducation, supportive psychotherapy, various group and individual therapies. Common components of these treatments involve (a) information about the disorder and its treatment; (b) practical support; (c) support for improving family communication; and (d) improving social and problem-solving skills and addressing maladaptive patterns of thinking about themselves and others<sup>6</sup>. The two most common structured psychological interventions are cognitive-behavioral therapy (CBT) and interpersonal therapy (IPT) that target maladaptive thoughts and behaviors using different techniques. A further psychological approach is psychodynamic psychotherapy (PDT) which is based on the principles of psychoanalysis. It aims to help patients increase awareness of their internal thoughts and patterns of behavior which might be contributing to their condition. Psychotherapy is considered a reasonable alternative to medication for mild depression and as an adjunct treatment in more severe depression where it can enhance response and reduce relapse <sup>7,8,9</sup>. However, psychological interventions require the active participation of patients as well as access to specialist therapies which might limit their real-world availability and efficacy.

# 8.1.3.3 Electroconvulsive Therapy (ECT)

Electroconvulsive therapy (ECT) is also referred to as electroshock or shock treatment mainly in the lay literature. During ECT, an electrical current is passed through the brain to produce an epileptic fit (otherwise known as convulsion or seizure). To minimize any discomfort, ECT is administered under general anesthesia. The current strength for ECT is usually around 800mA, which is 400 times higher than the current used for tDCS. Immediately after treatment, many patients experience headache, muscle aches and temporary amnesia about the period just prior to

<sup>&</sup>lt;sup>5</sup> Practice Guideline for the Treatment of Patients with Major Depressive Disorder. Third Edition, 2010. https://www.psychiatry.org/patients-families/depression/what-is-depression

<sup>&</sup>lt;sup>6</sup> National Alliance on Mental Illness. https://nami.org/About-Mental-Illness/Treatments/Psychosocial-Treatments

<sup>&</sup>lt;sup>7</sup> "Depression: The treatment and Management of depression in adults (updated edition)" Clinical guideline. NICE guidelines [CG90]. National Institute for Health and Care Excellence (UK). Published: October 2009, updated 2019. https://www.ncbi.nlm.nih.gov/books/NBK63748/pdf/Bookshelf NBK63748.pdf.

<sup>&</sup>lt;sup>8</sup> Practice Guideline for the Treatment of Patients with Major Depressive Disorder. Third Edition, 2010. https://www.psychiatry.org/patients-families/depression/what-is-depression

<sup>&</sup>lt;sup>9</sup> https://psychiatryonline.org/pb/assets/raw/sitewide/practice\_quidelines/quidelines/mdd.pdf



Protocol version: 9



the ECT. Confusion may also occur, mostly in elderly patients, that may last for up to 3 days (ref), and long-term memory dysfunction has been reported in patients. The ECT procedure was first conducted in 1938 and was initially used for a variety of mental health disorders conditions. Currently it is used mainly in patients with treatment-resistant depression. A meta-analysis on the effectiveness of ECT in MDD and bipolar depression conducted in 2012 reported overall remission rates of 51.5% for MDD and 50.9% bipolar depression. As of 2001, it was estimated that about one million people received ECT annually around the world.

# 8.1.3.4 Transcranial Magnetic Stimulation (TMS)

Transcranial magnetic stimulation (TMS) is a noninvasive procedure approved for the treatment of depression in Europe, Australia, and the US <sup>10</sup>. TMS is typically reserved for patients that have shown minimal or partial response to antidepressants and for patients for whom antidepressant treatment is not suitable. Each treatment session involves placing a purpose-made electromagnetic coil against the scalp in order to induce electric currents in the brain using repetitive magnetic pulses, hence the name repetitive TMS (rTMS). The treatment requires specialist equipment and medical supervision and is therefore not suitable for home use.

# 8.1.3.5 Cranial Electrotherapy Stimulation (CES)

Cranial electrotherapy stimulation (CES) (also referred to as cranial electrostimulation, electrosleep therapy, and electronarcosis) is a non-pharmacological, non-invasive treatment in which low-intensity electrical current is applied to the scalp. The main difference from tDCS is that CES uses alternating current (AC) rather than direct current (DC) electricity. There is currently a wide variety of CES devices. The Fisher Wallace Stimulator is a CES device which has FDA-approval for the treatment of anxiety, depression, and insomnia, and sold in the EU and Canada without a prescription, directly to consumers to be used at home.

#### 8.1.3.6 Transcranial Direct Current Stimulation (tDCS)

Flow is based on transcranial direct current stimulation (tDCS), a non-invasive brain stimulation technique where a weak direct current is applied on the scalp through electrodes. The current modulates the underlying neural activity. In principle, tDCS electrodes can be placed anywhere on the scalp. Changes in the tDCS electrode placement, also called montage, change the distribution of the induced electrical fields in the brain. Different montages are used depending on the indication. Empirical evidence indicates that a montage that targets the prefrontal cortex can reduce depression symptoms (see section 3.1.3 of the IDE (Attachment 001) for clinical data).

<sup>&</sup>lt;sup>10</sup> Carpenter LL, Janicak PG, Aaronson ST, et al. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of acute treatment outcomes in clinical practice. Depress Anxiety. 2012 Jul;29(7):587-96. doi: 10.1002/da.21969.



Protocol version: 9



#### 8.2 Investigational Device

#### 8.2.1 FLOW FL-100

Neuromodulation is a technique that alters neural activity through the targeted delivery of chemical or electrical stimulus. In particular, brain neuromodulation may be achieved through the direct application of stimulation via implanted deep brain stimulation (DBS) or non-invasively by TMS, CES or tDCS. Direct and non-invasive therapies have been tested for neurologic disorders such as Parkinson's disease, schizophrenia, chronic pain, and MDD, with MDD being the most studied disorder (Brunoni et al. 2010).

TMS to the dorsolateral prefrontal cortex (DLPFC) is shown in the literature to be safe and effective in treating MDD and as a result has received FDA clearance for MDD treatment (Cole et. al., 2019). TMS has proven to be commercially viable, however the treatment has some limitations. The limitations of TMS include the expensive capital equipment required for the delivery of treatment, which can only be delivered with specialist training. Patients being treated with TMS are required to attend multiple clinic visits, sometimes daily or multiple times daily, for weeks at a time, depending on their prescription.

Building from the understanding of the mechanisms, effects and targeting from TMS therapy, and removing some of the logistical hurdles that prevent access to TMS therapy, it is the intent of this study to investigate whether the area of the brain that is being modulated by TMS treatment can be similarly modulated by a home-use tDCS device, thereby offering a more affordable, accessible option for patients with MDD.

Flow Neuroscience has several years of experience developing and marketing tDCS devices for depression treatment. Its device, the Flow FL-100, is a CE-marked class IIa medical device for the treatment of Major Depressive Disorder (MDD). Flow FL-100 has been on the European market since mid-2019 and has been used by over 3000 patients. The product is currently available over the counter in the EU. Market approval has also been gained in Brazil.

Protocol version: 9





Figure 1. The Flow FL-100 Headset

The purpose of this trial is to investigate the use of the Flow FL-100 device to treat MDD at-home in a double-blind RCT.

#### 8.2.2 THE FLOW APP

The Flow app is used to control the Bluetooth connected Flow tDCS headset and acquire data about its use. The app is connected to a server that stores all data in a secure PostgreSQL database.

For the trial, a dedicated installation of the server and app will be used to isolate all trial data from data collected from retail Flow users. Trial participants will be given a link to the dedicated trial app (Google Play or Apple App store) before starting the trial. In the trial app, participants register with their email. No other identifying information is collected in the app. Only the Flow research team and Curebase will be able to log in to the Flow trial system and database and view the participant emails.

During the trial, the user will answer the nine questions of the MADRS-s form in the app. Answering the form is mandatory to continue with the stimulation. The app also continuously sends headset usage data to the server.

The trial personnel (at Curebase and at the sites in the UK and US) will have access to an administrative web interface where it can follow how much and when users have stimulated. This way they can monitor the usage of each patient and contact them if they start to miss sessions. This retention management is in addition to the normal Curebase retention management.





Figure 2. The Flow system and its components. A dedicated app and server will be used. Trial personnel will have access to an admin interface where they can view the activity of participants, unblind them, and move them to the open-label phase.



Figure 3 Flow trial admin interface - List of trial participants. Participants are identified through their email.

Protocol version: 9





Figure 4 Flow trial admin interface - View of an individual unblinded participant's data. Their MADRS-s scores and stimulation sessions are displayed. After unbinding the user's stimulation mode can be edited.

## 8.3 DEVICE TRACEABILITY

The US warehouse will maintain a Device Accountability Log to document the date of receipt, serial number, date of use, and final disposition of each device. The log will be available for review during monitoring visits. The Flow system also allows the trial personnel to see exactly which device has been used by which participant, and when.

Tracking of the investigational product used in this study will be consistent with 21 CFR Part 821 and ISO 14155:2020, and in accordance with local regulations. Devices will be stored in a secure location at the warehouses assigned for the trial (one in the US and one in Sweden).

At the end of the trial, all devices used in the US will be remotely disabled. Furthermore, a mechanism is in place to ensure that US trial devices cannot be used in the customer-facing Flow app. UK participants will be allowed to keep their devices.

Protocol version: 9



#### 8.4 Supply and Accountability of Investigational Devices

The full name and address are needed for shipping the devices to the participants' homes. There will be one warehouse in Sweden and one in the US. The warehouse in Sweden is the same as used for normal Flow customers, and the warehouse in the US will be dedicated to the trial. To ensure that only limited personnel at Flow have access to shipping information, special accounts in the shipping partners' software systems will be set up. This will isolate information from the normal operations of Flow. Only the CTO from Flow Neuroscience will be able to access the shipping information of participants.

The sponsor is: Flow Neuroscience AB Södra Förstadsgatan 2 211 43 Malmö

Tele: +46736607170

erik@flowneuroscience.com

#### 8.5 Device Use Experience and Training

The study Sponsor will ensure appropriate training for each investigator prior to initiation of the study at each investigational site. Investigators will be trained on the Flow FL-100 device by the Sponsor, and/or qualified representatives of the Flow FL-100 device prior to their participant's first use. This training will address topics such as the indications and contraindications for the use of the device, device handling, instructions for use and device instrumentation.

In addition, the Sponsor will provide training on the protocol, participant selection criteria, AE management, and follow-up.

## 9 Benefit-Risk Analysis

#### 9.1 RISKS

The study device will deliver a maximum of 2 mA tDCS for 30 minutes at a time. Published data has shown conventional sessions to be  $\leq$  40 minutes at  $\leq$  4mA, and the tolerability and dropout rates between sham and active stimulation groups are equal in the literature.

As of August 2021, the most common side effects reported in the literature and from post-market data on Flow FL-100 are:

Table 4. Common side effects from Flow FL-100

| Side Effect | % of users |
|--------------------------|------------|
| Skin irritation, redness | 0.80% |

Protocol version: 9



| Strong tingling, stinging, or itching | 0.14% |
|---------------------------------------|-------|
| Headache | 1.1% |
| Increased tinnitus | 0.45% |

Most people also experience skin redness at the stimulation site which passes within 30 minutes after the stimulation. Small skin burns are also known from the literature due to the use of tap water instead of physiological saline to wet the stimulation electrodes<sup>11</sup>. Therefore, Flow is delivered with disposable pre-moistened sponges so that the users do not need to handle saline themselves.

The tDCS studies in participants with MDD have reported mostly consistent adverse events with large studies on healthy participants<sup>12</sup>. In addition to this, there have been four studies that have published the appearance of treatment-emergent mania/hypomania (TEM) in eleven cases total<sup>13</sup>. Most cases of TEM have been where tDCS has been combined with antidepressant drugs, which are known to increase the risk of a manic switch<sup>14</sup>. As such, a causal relationship has not been determined. The observed cases have also been mild and in general not required any intervention (correspondence with authors). In the internal data from over 3,000 Flow FL-100 users, no instance of TEM has been discovered or reported. In accordance with the recommendation from Antal et al. (2017), participants with a history of bipolar disorder will be excluded from this study due to their increased risk of manic switch. As an additional safety measure, the YMRS will be administered at each follow-up visit.

#### 9.2 RISK MITIGATION

An evaluation of the potential risks associated with use of the Flow FL-100 device has been performed to minimize the risks associated with the device. The following are some of the ways in which risks have been or will be minimized:

<sup>&</sup>lt;sup>11</sup> Palm U, Keeser D, Schiller C, et al. Skin lesions after treatment with transcranial direct current stimulation. Brain Stimul 2008;1:386e7. [7] Frank E, Wilfurth S, Landgrebe M, et al. Anodal skin lesions after treatment with transcranial direct current stimulation. Brain Stimul 2010;3:58e9.

<sup>&</sup>lt;sup>12</sup> Antal A, Alekseichuk I, Bikson M, Brockmöller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Flöel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID: 28709880; PMCID: PMC5985830.

<sup>&</sup>lt;sup>13</sup> André R. Brunoni, Adriano H. Moffa, Bernardo Sampaio-Júnior, Verònica Gálvez, & Colleen K. Loo (2017). Treatment-emergent mania/hypomania during antidepressant treatment with transcranial direct current stimulation (tDCS): A systematic review and meta-analysis. *Brain Stimulation*, 10(2), 260-262.

<sup>&</sup>lt;sup>14</sup> Patel R, Reiss P, Shetty H, Broadbent M, Stewart R, McGuire P, Taylor M. Do antidepressants increase the risk of mania and bipolar disorder in people with depression? A retrospective electronic case register cohort study. BMJ Open. 2015 Dec 14;5(12):e008341. doi: 10.1136/bmjopen-2015-008341. PMID: 26667012; PMCID: PMC4679886.

Protocol version: 9



#### 9.2.1 Monitors

All Flow devices are controlled by the app and the app is connected to the Flow server over the internet. It is possible to disable devices remotely; this feature ensures patient safety in case of malfunction. This feature is not available for other tDCS devices. The frequency of use of each individual Flow device is remotely monitored and therefore it is possible to assess adherence to treatment. We expect the Flow device to enhance patient clinical care in general, given the ability for physicians to have remote access to real-time patient data.

#### 9.2.2 Stimulation Parameter Space

Stimulation will always have a maximum output of 2 mA.

#### 9.2.3 Usage Limits

Since Flow is controlled by the accompanying app it limits how often the device can be used and therefore this risk is mitigated. The treatment protocol is however the same for both devices with up to 5 sessions per week the first 3 weeks and then 3 sessions per week. With a maximum of one 30-minute session per day.

#### 9.3 ANTICIPATED BENEFITS

Participants may experience a clinically meaningful improvement in MDD as has been shown in previous placebo controlled clinical studies with similar therapy. Based on the self-reporting Flow FL-100 users complete every week, over 80% report having some improvement in their depression and around 30% reach remission in 6 weeks. It is also possible that participants will not experience a clinical benefit from participation, although there may be a beneficial addition to the body of knowledge for this therapy. There may be benefits that are unforeseen at this time. Flow also gives participants access to a type of treatment that is in general only available at clinics.

The remission rate of 30% is consistent with what has been found in the literature on tDCS for depression treatment using other devices.

#### 9.4 RISK-TO-BENEFIT RATIO

All applicable risks have been addressed through appropriate testing and clinical monitoring. Any residual risks are acceptable when weighed against the potential benefits to the participant. The device is appropriate for the intended use and is designed to protect the health and safety of the participant, user, and environment.

Therefore, the risk/benefit profile of the Flow FL-100 in the intended use justifies the conduct of the proposed clinical investigation.

#### 10 Study Objectives

#### 10.1 BACKGROUND

To conduct a double-blind, placebo-controlled, randomized, superiority, remote trial for individuals with major depressive disorder.

Protocol version: 9



#### 10.2 PRIMARY OBJECTIVE

To show that active stimulation with the Flow FL-100 device is superior to sham stimulation for the treatment of major depressive disorder when used at-home.

#### 11 STUDY DESIGN

The study will be lead by Professor of Affective Neuroscience Cynthia Fu, PhD, MD, University East London (UK site) and Associate Professor of Psychiatry Sudhakar Selvaraj, PhD, MD, University of Texas Health Sciences center at Houston (UTHealth) (US site), both with extensive experience in managing clinical trials and treating MDD. The other co-investigators are Dr. Jair Soares, PhD, MD, Chairman and Professor of Psychiatry at UTHealth, Houston and Dr. Marsal Sanches, PhD, MD, Associate Professor of Psychiatry at UTHealth, Houston, both have a long history of leading and managing clinical trials and treating MDD and Psychiatric disorders. The other study site investigators are well trained researchers with graduate or postgraduate degrees with training and experience in clinical studies. The study Pls and Co-ls will provide day-to-day supervision to the study investigators and responsible for the overall conduct of the study.

#### 11.1 STUDY DURATION

The study is expected to take approximately 10 months from first participant enrolled to the last open-label visit.

- 5 months enrollment period (estimation)
- 5 months treatment and open-label

The follow-up period during the clinical investigation shall permit the demonstration of performance over a period, sufficient to represent a realistic test of the performance of the investigational device and allow any risks associated with adverse device effects over that period to be identified and assessed.

#### 11.2 TREATMENT/CONTROL GROUPS

For each participant, the trial will be conducted in 2 phases: blinded and open label.

Protocol version: 9





Figure 5 Participant Activity Flowchart

#### 11.3 BLINDED PHASE

During the treatment phase, the participants will be randomized into one of the two arms: active and sham. The participants will be divided equally between the arms and will not be informed of their assignment. The participants will be informed during the consent process that some of them will have sham stimulation during their initial 10-week participation, depending on their randomization assignment.

The sham group receives sham stimulation following how sham tDCS is normally implemented in clinical trials. At the beginning of each 30-minute stimulation session, the current is ramped up to 1mA over 30 seconds. However, when it has reached its maximum, it is again slowly ramped down to 0 mA over 15 seconds. By the end of the session, the current is then again ramped up to 1 mA over 30 seconds and then ramped down to 0 mA over 15 seconds.

The 1 mA current, compared to 2 mA for active stimulation, allows the user to feel the tingling of the stimulation but while still minimizing the amount of current they are exposed to.

When in sham, the app user interface behaves exactly as if the stimulation was active. This way the participants will be blind to the mode of stimulation. If for some reason the stimulation is paused during stimulation the same ramp up and down procedure is done again when the stimulation is resumed.

Protocol version: 9





After the trial period, all user's devices will start working, and users who received sham stimulation can choose to restart the treatment with active stimulation.

# 11.4 OPEN LABEL PHASE

After the completion of the blinded treatment phase all participants will be offered to continue the treatment. Members of the sham group will be offered to restart the treatment with active stimulation, while members of the active group will be offered to continue maintenance treatment for 10 more weeks at 3 sessions per week.

#### 11.5 PRIMARY ENDPOINTS

The primary effectiveness endpoint is the adjusted mean group difference in the HDRS-17 scores at 10 weeks compared to baseline for subjects in the Active device and the Sham device groups.

#### 11.6 SECONDARY ENDPOINTS

- Arm difference in HDRS-17 response and remission rate at week 10.
- Arm difference in MADRS average score change, and response and remission rate at week 10.
- Arm difference in MADRS-s average score change, and response and remission rate at week 10.
- Quality of life improvement as measured by EQ-5D-3L in the active compared to sham arm at week 10.

#### 11.7 EXPLORATORY ENDPOINTS

- Young Mania Rating Scale (YMRS) at 10 weeks.
- tDCS Adverse Events Questionnaire (AEQ) at 10 and 20 weeks
- Hamilton Anxiety Rating Scale (HAM-A) change at week 10.



Protocol version: 9



- HDRS-17, MADRS, MADRS-s mean decrease, and remission and response rate at 20 weeks (after open-label) compared to open-label start and baseline.
- Correlation between MADRS and MADRS-s.
- Correlation between adherence to stimulation and HDRS-17/MADRS decrease in the active group at 10 weeks.
- Neuropsychological measure: verbal learning (Rey Auditory Verbal Learning Test (RAVLT) and information processing speed (Symbol-Digit Modalities Test (SDMT)
- Treatment acceptability questionnaire (TAQ) as developed by UEL. There is one form at baseline and another at week 10 and 20.
- The within-patient clinically meaningful improvement as defined as at least -3 points on the HDRS-17 scale. The percentage of subjects for each arm that reaches -3 points or more improvement and also the Cumulative Distribution Function Curves of Change in HDRS-17 Score from Baseline to Primary end-point by arm.

#### 12 Selection of Study Population

#### 12.1 Participant Recruitment

Participants in this study will be recruited via the Flow Neuroscience website, email lists, and online marketing. Potential participants will be directed to a pres-creening form hosted by Curebase, they will then be required to sign up/register with the Curebase platform to complete a pre-screening survey. This information will primarily be used to screen potential participants for eligibility. Users will be given general information about the trial, and that is it will be blinded.

Participants who seem to meet preliminary eligibility will have a virtual pre-screening visit with a Curebase coordinator prior to being sent to a site investigator for informed consent and further screening procedures. Participants must meet all the following inclusion criteria and none of the exclusion criteria. The investigator maintains exclusive responsibility for the inclusion and exclusion of any potential study participant.

#### 12.2 INCLUSION CRITERIA

To be eligible to participate in this study, participants must meet all the following criteria:

- 1. Be ≥18 years.
- Have a diagnosis of Unipolar MDD with a current depressive episode as defined by the diagnostic criteria in the Diagnostic and statistical manual of mental disorders – 5th edition (DSM-V
- 3. Have a Hamilton Depression Rating Score (HDRS-17) of ≥ 16.
- 4. For 6 weeks prior to enrollment, are either:
  - a. not taking antidepressant medication or:

Protocol version: 9



- b. are taking a stable antidepressant regimen with a stable medication source and agree to continue the same regimen throughout study participation
- 5. If in psychotherapy, have maintained stable psychotherapy for at least 6 weeks prior to enrollment.
- 6. Have access to a stable internet connection through which the treatment will be received.
- 7. Have access to a smartphone or other device running Android 5.0+ or iPhone Operating System (iOS) 12+ (e.g., reasonably new iPhone/iPad or Android phone), used to using the device in their everyday life, and can capably use the study application on the device, as determined by the investigator.
- 8. Are currently living in England/Wales (UK) or Texas (US).
- 9. Subject is currently under the care of a psychiatrist or a primary care physician, agrees to be evaluated at regular intervals by a psychiatrist or primary care physician for the duration of study participation, and agrees to promptly inform the study staff of any change of psychiatric or mental health providers during study participation.
- 10. Subject agrees to allow any and all forms of communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within at least two years of study enrollment.
- 11. Subject agrees to provide the name and verifiable contact information (email and mailing addresses, mobile and land-line phone numbers, as applicable) of at least two persons ≥ age 18 who reside within a 60-minute drive of the patient's residence and whom the research staff is at liberty to contact, as they deem necessary, for the duration of study participation.
- 12. Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study.
- 13. Be willing and able to comply with all study procedures.
- 14. Subject agrees to meet all of the inclusion criteria throughout their participation in the study. Otherwise, the subject will be discontinued from the study.
- 15. Subject agrees to a Safety/Suicide Risk Management Protocol, which is intended to reduce the reduce the risk of suicide during study participation.

#### 12.3 Exclusion Criteria

Participants who meet any of the following criteria will be excluded from participating in this study:

- 1. Are in a current state of mania, as determined by the YMRS or psychosis, as determined by the MINI.
- 2. Are diagnosed with vitamin or hormonal deficiencies that may mimic mood disorders, as determined by the investigator.
- 3. Are currently receiving any other interventional therapy for MDD other than a stable regimen of antidepressants or psychotherapy as defined in the inclusion criteria.
- 4. Considered to have treatment resistant depression as defined by inadequate clinical response to 2 or more trials of antidepressants at an adequate dose and duration.
Protocol version: 9



- 5. Have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), cranial electrotherapy stimulation (CES), transcranial direct current stimulation (tDCS), deep brain stimulation (DBS), or other brain stimulation.
- 6. Patient answers Yes to Questions 4, 5 or 6 on the Columbia Suicide Severity Rating Scale (C-SSRS) Triage and Risk Identification Screener.
- 7. Any previous hospitilization for suicidal behavior.
- 8. Have chronic severe insomnia (< 4 hours of sleep each night), or depression secondary to chronic insomnia or sleep apnea
- 9. Have any structural lesion (e.g., any structural neurological condition, or more subcortical lesions than would be expected for age or have had a stroke that affects stimulated area or connected areas) or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results, as determined by the investigator.
- 10. Have any implant in the brain (e.g., DBS) or neurocranium, or any other active implantable medical device.
- 11. Have any neurocranial defect.
- 12. Have a history of epilepsy or seizures (including history of withdrawal / provoked seizures).
- 13. Have shrapnel or any ferromagnetic material in the head.
- 14. Have any disorder that would impair the ability to complete the study questionnaires.
- 15. Have been diagnosed with autism spectrum disorder.
- 16. Are actively abusing substances (<1 week prior to enrollment).
- 17. Have a cognitive impairment (including dementia).
- 18. Have a history of mania or psychosis.
- 19. Are currently using any medications that affect cortical excitability (e.g., benzodiazepines, epileptics, etc.).
- 20. Are currently experiencing symptoms of withdrawal from alcohol or benzodiazepines.
- 21. Have been diagnosed with Parkinsonism or other movement disorder as determined by the investigator to interfere with treatment.
- 22. Have ever taken esketamine / ketamine for treatment of depression.
- 23. Have ever been admitted to hospital for depression.
- 24. Have ever been diagnosed with obsessive-compulsive disorder (OCD) or bipolar type 1 or 2 disorder.
- 25. Is diagnosed with an active primary anxiety disorder, or PTSD, agoraphobia, anorexia or bulimia, panic or personality disorder with active symptoms.
- 26. Have a history of psychosurgery for depression.
- 27. Have any history of myocardial infarction, coronary artery bypass graft (CABG), coronary heart failure (CHF), or history of other cardiac issues.
- 28. Are currently experiencing or have a history of intractable migraines.
- 29. Are a chronic tobacco smoker, as defined by smoking by smoking >100 cigarettes (including hand-rolled cigarettes, cigars, cigarillos, etc.) in their life-time and have smoked every day for the last 7 days.



Protocol version: 9



- 30. If female and of child-bearing potential, currently pregnant or breastfeeding or planning to become pregnant or breastfeed any time during the study.
- 31. Are currently a prisoner.
- 32. Are participating concurrently in another clinical investigation or have participated in a clinical investigation within the last 90 days or intend to Participate in another clinical investigation during the study, and where the participation in the other investigation might interfere with the results of this trial as deemed by the PI.
- 33. Have any medical condition or other circumstances, in the judgment of the investigator, that might interfere with the ability to complete follow-up visits and the self-reported MADRS-s in the app.
- 34. Have any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the device's safety and performance.
- 35. A Subject who meets any of the exclusion criteria during study participation will be discontinued from the study

# 12.4 Study Enrollment Procedures

All participants with MDD will be considered for screening into the study. Participants expressing an interest in participation will proceed with the consent process as per section 13.1 Informed Consent. A participant is not considered officially enrolled in the study until after signing the study consent form.

#### 12.4.1 Participant Enrollment

Participants who consent to participate shall be assigned a unique Participant Identification Number to de-identify their information. This Participant Identification Number will be captured in the Curebase platform and used to identify them on all source documents and eCRFs thereafter.

A record of all screened participants will be maintained in the Curebase platform. The date of screening, results of screening (included or not) and, if not eligible, the primary reason for excluding the participant, enrollment status (enrolled or not) and, if not enrolled, the primary reason will be recorded.

Please note, for purposes of the study a participant is considered enrolled at informed consent.

NOTE: If a participant does not meet the eligibility criteria during their initial screening, the participant cannot be re-evaluated for entry into the study later.

# 12.5 SCREEN FAILURES

A screen failure participant is a consented participant that did not receive the Flow FL-100 treatment due to withdrawing consent, being withdrawn from the study, or not meeting eligibility requirements for treatment.



Protocol version: 9



If a participant signs the ICF but is found ineligible for inclusion in the study prior to receiving the Flow FL-100, the participant will not be advanced any further in this clinical investigation. The participant's signed ICF and completed inclusion/exclusion criteria will be retained by the Investigator, and the participant will be notified.

Screening data from the Screening Visit including the reason for exclusion, will be collected but may not be complete in cases where the participant is determined to be a screen failure early in the screening process. The participant's exclusion from the study, and reason for ineligibility, will be documented in the Screening & Enrollment Log.

#### 12.6 Participant Treatment Assignment

During the technical onboarding session at Week 0, the participant will receive the link to the app and a code to access the app. The participant will download the app and sign up in the app with their email, password, and app access code. When the participant creates their account in the trial app they will automatically be randomized to the sham or active treatment arm (with 50% probability). Block randomization is used with randomly permuted block sizes of 4 and 6. This is done by the trial server and stored in its dedicated database. No one who is working with the trial will have access to the raw data until it has ended.

## 13 Study Procedures

# 13.1 WEEK -3 TO -1: INFORMED CONSENT (ICF)

After passing the screener survey, prospective participants will be directed to review and sign an electronic HIPAA, and an IRB/EC-approved consent (eConsent) form that are hosted in the Curebase system. The eConsent form will explain the nature and scope of the study, the procedures to be performed as part of the study, the potential risks, and benefits of participation, expected duration of participation, possible treatment alternatives, and an overview of his/her rights as a study participant in lay terms. Participants will have the opportunity to discuss the study with their family or surrogates or think about it before agreeing to participate. Participants will be informed that participation is voluntary and will be assured that they may withdraw from the study at any time and for any reason, without repercussion.

After viewing the eConsent materials, participants will have an opportunity to email or call the research team with any questions they may have and will be given as much time as needed to receive answers before making a final decision regarding study participation. Participants will receive a telephone number, email, and will have access to contact support staff as needed.

When the individual is ready to confirm their willingness to participate, an electronic signature will be collected to complete the eConsent formalities. The participant will receive a copy of the fully signed HIPAA, and eConsent forms via email to retain for their records, and a digital copy will be retained within the Curebase system as part of the study records.

Upon successful documentation of informed consent, a screening video call will be performed and will serve as a baseline evaluation to confirm patient eligibility.

Protocol version: 9



- Clinician Reported Outcome (ClinRO)
  - Hamilton Depression Rating Score (HDRS-17)
  - Montgomery–Åsberg Depression Rating Scale (MADRS)
  - Mini International Neuropsychiatric Interview (MINI)
  - Hamilton Anxiety Rating Scale (HAM-A)
  - Young Mania Rating Scale (YMRS)
  - Rey Auditory Verbal Learning Test (RAVLT)
- Patient Reported Outcome (PRO) Questionnaires
  - EQ-5D-3L
  - Symbol-Digit Modalities Test (SDMT)
  - Treatment Acceptability Questionnaire (TAQ)
  - tDCS Adverse Events Questionnaire (AEQ)
  - Columbia Suicide Severity Rating Scale (C-SSRS)
- Review of concomitant medications
- Final review of inclusion/exclusion criteria
- Intervention kit will be shipped to the participant

# 13.2 WEEK 0

To allow the Investigator's assessment of the participant's progress, the participant will complete a video call with study staff and undergo the following:

- Review of concomitant medications
- Record any new or updated adverse events and device deficiencies, if applicable
- SDMT baseline
- Technical onboarding & device training session
- Randomization

## 13.3 WEEKS 1, 4 & 7

To allow the Investigator's assessment of the participant's progress, the participant will complete a video call with study staff and undergo the following:

- ClinROs
  - HDRS-17

Protocol version: 9



- MADRS
- YMRS
- C-SSRS
- Review of concomitant medications
- Record any new or updated adverse events and device deficiencies, if applicable

#### 13.4 WEEK 10

To allow the Investigator's assessment of the participant's progress, the participant will complete a video call with study staff and undergo the following:

- ClinROs/PROs
  - HDRS-17
  - MADRS
  - HAM-A
  - YMRS
  - EQ-5D-3L
  - RAVLT
  - SDMT
  - TAQ
  - AEQ
  - C-SSRS
- Review of concomitant medications
- Record any new or updated adverse events and device deficiencies, if applicable

For participants in the Sham Arm:

 Participants in the Sham arm will be informed of their assignment and will be offered to start active, Open-Label stimulation for 10 weeks, with 5 sessions the first 3 weeks and then up to 3 sessions per week.

For participants in the Active stimulation Arm:

• Participants in the Active arm will be offered to continue maintenance treatment for 10 more weeks at 3 sessions per week.

13.5 WEEK 20 FOLLOW-UP VISIT - OPEN-LABEL ONLY

To allow the Investigator's assessment of the participant's progress, the participant will complete a video call with study staff and undergo the following:



Protocol version: 9



- ClinROs/PROs
  - HDRS-17
  - MADRS
  - HAM-A
  - YMRS
  - EQ-5D-3L
  - RAVLT
  - SDMT
  - TAQ
  - AEQ
  - C-SSRS
- Review of concomitant medications
- Record any new or updated adverse events and device deficiencies, if applicable.

## 13.6 VIDEO CALLS

All trial visits will be conducted remotely using real-time video conferencing.

The site personnel who will conduct remote visits will be trained on how to conduct real-time video conferencing visits (e.g., trained on the use of telemedicine for remote clinical trial visits).

Both the researcher and the trial participant should confirm their respective identities with one another before engaging in a visit by showing a photo ID to the camera.

The date and time of a visit should be documented in the trial records.

#### 13.7 LATE AND MISSED VISITS

If a participant fails to return for a scheduled study visit within the visit window defined in the study protocol but completes the visit prior to the beginning of the next visit window, that visit is considered to have been completed late. A protocol deviation should be documented on the appropriate eCRF.

If a participant fails to return for a scheduled study visit within the visit window defined in the study protocol and the next scheduled study visit window opens, that visit is considered to have been missed. A protocol deviation should be documented on the appropriate eCRF.

Protocol version: 9



All attempts should be made to schedule the participant for the study visit as soon as possible so that it is captured late rather than missed completely.

## 13.8 Unscheduled Visits

Participants may be seen for unscheduled visits as needed. During the unscheduled visit, the Investigator will assess the participant's progress and perform the following:

- ClinROs
  - HDRS-17
  - MADRS
  - YMRS
  - C-SSRS
- Review of concomitant medications
- Record any new or updated adverse events and device deficiencies, if applicable

## 13.9 Study Completion/Discontinuation

The Primary Endpoints will be evaluated at 10 weeks. Participants will complete study participation at 10 weeks unless consented and enrolled in an additional 10-week open-label portion of the study. Participants enrolled in the open-label phase will complete the trial after 20-weeks.

## 14 Description of Study Procedures

#### DEMOGRAPHICS

At screening, participant baseline characteristics including, but not limited to, age and gender, will be recorded.

## PAST MEDICAL HISTORY

At screening, each participant's past medical conditions and surgical procedures will be recorded.

#### Pregnancy Determination

Prior to treatment, female participants of childbearing potential will be asked during the Screening visit whether they are pregnant or breastfeeding or plan to become pregnant or breastfeed during the trial.

## CLINICIAN AND PATIENT REPORTED OUTCOME QUESTIONNAIRES (CLINROS/PROS)

The following Clinician or Patient Reported Outcome questionnaires will be completed and used to compare participant outcomes at follow-up time points compared to baseline:

Montgomery-Asberg Depression Rating Scale (MADRS) - ClinRO



Protocol version: 9



The Montgomery–Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.

# Montgomery-Asberg Depression Rating Scale (MADRS-s) - PRO

MADRS-s is a self-rating version of MADRS and correlates well with expert ratings. The MADRS-s instrument has nine questions, with an overall score ranging from 0 to 54 points. During the trial, each participant reports their MADRS-s score in the same way as normal customers would. The MADRS-s uses cut-off points detailed below to classify the severity of depressive symptoms:

• 0-12 points: None or very mild depression

• 13-19 points: Mild depression

• 20-34 points: Moderate depression

• ≥ 35 points: Severe depression

# Hamilton Depression Rating Score (HDRS-17)

The HDRS (also known as the Ham-D) is the most widely used clinician-administered depression assessment scale. The original version contains 17 items pertaining to symptoms of depression experienced over the past week. The questionnaire is designed to be used by clinicians to rate the severity of depressive symptoms in adults by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms.

# Mini International Neuropsychiatric Interview (MINI) - ClinRO

The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a short structured diagnostic interview, developed jointly by psychiatrists and clinicians in the United States and Europe, for DSM-IV and ICD-10 psychiatric disorders.

# Columbia Suicide Severity Rating Scale (C-SSRS) - ClinRo

The Columbia Suicide Severity Rating Scale, or C-SSRS, is a rating scale to evaluate suicide risk. The scale identifies specific behaviors which may be indicative of an individual's intent to kill oneself.

#### Hamilton Anxiety Rating Scale (HAM-A) - ClinRo

The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms and is still widely used today in both clinical and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).



Protocol version: 9



# Young Mania Rating Scale (YMRS) - ClinRo

The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours.

# Rey Auditory Verbal Learning Test (RAVLT) - ClinRo

The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological assessment designed to evaluate verbal memory in patients, 16 years of age and older. The RAVLT can be used to evaluate the nature and severity of memory dysfunction and to track changes in memory function over time.

## Symbol-Digit Modalities Test (SDMT) - PRO

The Symbol Digit Modalities Test (SDMT) detects cognitive impairment. It is a way for clinicians to screen for organic cerebral dysfunction in both children (eight years and older) and adults. The SDMT is brief, easy to administer, and has demonstrated sensitivity in detecting not only the presence of brain damage, but also changes in cognitive functioning over time and in response to treatment.

## Treatment Acceptability Questionnaire (TAQ) - PRO

TAQ is a questionnaire for probing how acceptable participants of tDCS clinical trial think the treatment is. At baseline it measures participant's expectations about the trial, e.g., treatment outcome, effort needed, ethics, etc., and then follow-up on these expectations at the end of the trial.

## tDCS Adverse Events Questionnaire (AEQ) - PRO

AEQ is a specialized questionnaire developed to capture the adverse events during tDCS trials.

## EQ-5D-3L - PRO

The EQ-5D-3L is a standardized measure of health-related quality of life.

# 15 EARLY DISCONTINUATION: PARTICIPANTS

## 15.1 TECHNICAL FAILURES

In case the Flow device or the participant's smartphone breaks, and it cannot be replaced within 10 days, and the participant has not already completed 22 sessions, this will be considered a technical failure, and the participant will be withdrawn from the trial.

## 15.2 Treatment Failures

The following situations will be considered treatment failures and participants will be withdrawn from the trial:



Protocol version: 9



- 30% increase in HDRS-17 score compared to baseline.
- Suicidal attempts / completion
- Device related SAE

# 15.3 Lost to Follow-Up (LTFU)

Participants who miss the final, 10-week study visit will be regarded as Lost to Follow-Up. As described in the Statistical Analysis Plan, these subjects will be included in the primary analysis through Multiple Imputation. Therefore, this definition of LTF only applies to study operations and not data analysis. Curebase or site staff should perform and document a minimum of three attempts to contact them via phone to complete the final study visit prior to considering the participant LTFU. The Curebase or site staff should document the date and type of attempted communication.

All efforts should be made to have participants complete all follow-up visits.

#### 15.4 WITHDRAWALS

Participants have the right to withdraw from the clinical investigation at any time and for any reason. The Principal Investigator will ask the reason for their withdrawal and will record all information regarding the participant discontinuation.

A Participant may be withdrawn from the clinical investigation for the following reasons:

- Participants may choose to withdraw from the clinical investigation under the terms of the Declaration of Helsinki and their consent documentation without having to give a reason;
- Any unanticipated adverse event which, in the opinion of the Principal Investigator, is related to the treatment and will endanger the well-being of the participant if treatment is continued:
- Development of any intercurrent illness(es), infection or condition(s) that might interfere with the clinical investigation;
- Non-compliance with the clinical investigation procedures deemed by the Principal Investigator to be sufficient to cause discontinuation;
- Any problem deemed by the Investigator to be sufficient to cause discontinuation.

Participants will be withdrawn from the trial if they do not comply with the intervention, namely if they are unable to have a minimum of 60% of the tDCS session (22 (660 minutes) out of 36 sessions at week 10) during the blinded phase, or if they develop serious adverse effects from any part of the study. Recording of the reasons for withdrawal will be made. Their GP will be informed about their withdrawal, and they will have a telephone follow up at 1 month following their withdrawal.

If a participant is withdrawn, their device is disabled to make sure they cannot continue the treatment.



Protocol version: 9



Regardless of the reason for withdrawal, data available for the participant at the time of withdrawal, including the reason for withdrawal, will be entered on the Case Report Forms. The research staff will request to have an optional early termination visit to collect the same data as at the week 10 and week 20 interview. The Principal Investigator will treat all participants discontinued from the investigation due to an unanticipated adverse event, directly related to the investigation, until the reaction resolves. A participant that has been withdrawn from the study after treatment start will not be replaced.

#### 15.5 DOCUMENTATION OF EARLY DISCONTINUATION AND PREGNANCY

In every instance where a participant does not complete the study, the Investigator will document the primary reason for discontinuation in the participant's records.

All participants are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. However, if a participant expresses a desire to withdraw their consent for the study, the site should attempt to obtain written documentation for their study records.

For participants that are discontinued by the Investigator, the Investigator must notify them of their discontinuation from the study in writing.

To ensure the safety of participants who become pregnant during the study, pregnant participants will be withdrawn from the study.

## 15.6 Use of Data from Early Discontinuation Cases

Study data collected previously for participants who withdraw from the study, are discontinued from the study by the Investigator or LTFU will be included in the data analysis and clinical study report.

15.7 Ongoing Treatment for Early Discontinuation Cases

Participants who withdraw voluntarily or are discontinued by the Investigator will remain eligible for SOC treatment by the Investigator and study staff.

- 16 Early Discontinuation: Study
- 16.1 Procedure for Suspension or Early Termination

The Sponsor may suspend or prematurely terminate this clinical investigation either at an individual investigational site or at all sites. A Principal Investigator, IRB/EC, or regulatory authority may suspend or prematurely terminate participation in this clinical investigation at the investigational sites for which they are responsible.

If suspicion of an unacceptable risk to participants arises during the clinical investigation, or when so instructed by the IRB/EC or regulatory authorities, the Sponsor will suspend the clinical



Protocol version: 9



investigation while the risk is assessed. If an unacceptable risk is confirmed, the Sponsor will terminate the clinical investigation.

The Sponsor will consider terminating or suspending the participation of a particular investigational site or Investigator if monitoring or auditing identifies serious or repeated deviations on the part of an Investigator.

If suspension or premature termination occurs, the terminating party will justify its decision in writing and promptly inform the other parties with whom they are in direct communication.

If suspension or premature termination occurs:

The Sponsor will remain responsible for providing resources to fulfill the obligations from this protocol and existing agreements for following the participants enrolled in the clinical investigation, and the site's Principal Investigator or authorized designee will promptly inform the enrolled participants at his/her investigational site

If the study is terminated, Flow Neuroscience AB must comply with all applicable government regulations and the protocol-required participant follow-up. If discontinuation of the study should occur, the Principal Investigator must return all clinical investigation materials (including devices) to the Sponsor and provide a written statement to the IRB/EC explaining the reasons for the premature termination. All applicable clinical investigation documents shall be participant to the same retention policies, as detailed in Section 24.3.

## 16.2 Procedure for Resuming the Clinical Investigation After Temporary Suspension

When the Sponsor concludes an analysis of the reason(s) for the suspension, implements the necessary corrective actions, and decides to lift the temporary suspension, the Sponsor will inform the relevant parties of the rationale and provide them with the relevant data supporting this decision. Concurrence will be obtained from the IRB/ECs and, where appropriate, regulatory authorities before the clinical investigation resumes. If participants have been informed of the suspension, the Principal Investigator or authorized designee will inform them of the reasons for resumption.

### 16.3 ROUTINE CLOSE-OUT

Routine close-out activities will be conducted to ensure that the Principal Investigator's records are complete, all documents needed for the Sponsor's files are retrieved, remaining clinical investigation materials are destroyed, previously identified issues have been resolved, and all parties are notified.

## 17 Protocol Deviations

Conformance to the protocol is essential to the quality and integrity of the clinical study. Every effort should be made to avoid any deviation from the clinical protocol. A protocol deviation is an event



Protocol version: 9



whereby the clinical investigator or site personnel did not conduct the study according to the protocol.

Under emergency circumstances, deviations from the protocol to protect the rights, safety and well-being of human subjects may proceed without prior approval of the sponsor and the IRB/EC. Such deviations shall be documented and reported to the sponsor in the EDC within 5 days of knowledge. The IRB/EC should be notified of the deviation as required by IRB/EC reporting guidance.

### 18 CONCOMITANT MEDICATIONS/THERAPIES

For the purposes of this clinical study, only medications taken or administered for the following will be recorded (*Ensure medications reflected in incl/excl are listed here*):

- Muscle relaxation;
- Other medications related to or given for the participant's MDD.

# 19 Adverse Event & Device Deficiency Reporting

Subjects will be carefully monitored during the study for possible adverse events (AEs) from the time they sign the Informed Consent Form to the time of study completion. All medical events and conditions prior to this time point are to be captured as medical history.

Any observed unanticipated AE will be fully investigated by the Investigator and classified in line with the definitions of ISO 14155:2020 below. The frequency and severity of anticipated AEs will instead be captured using the tDCS Adverse Events Questionnaire (AEQ).

All unanticipated adverse events that occur during this study will be recorded on the adverse event eCRFs and must include the following information at minimum:

- Event Description
- Date of Onset
- Date of Resolution
- Severity
- Seriousness
- Relationship to Study Device/Procedure
- Outcome

Adverse events will be reported and classified by the Investigator using the specific signs, symptoms or abnormal laboratory values, or medical diagnosis if no signs, symptoms, or abnormal laboratory values can be identified.

Protocol version: 9



Significant new information and updates should continue to be captured in the subject's records and in the EDC as they become available and the adverse event should be followed until it is resolved or no further improvement is expected, or the subject is lost to follow-up.

Adverse events that meet the definitions of seriousness in Section 19.1 below should also be reported to the Sponsor per the instructions provided in Section 19.2.4 below.

# 19.1 Definitions

The following definitions are from the ISO 14155:2020 and MDCG 2020-10:

**Adverse Event (AE)** – An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings.) in subjects, users, or other persons, whether or not related to the investigational device and whether anticipated or unanticipated.

NOTE 1: This definition includes events related to the investigational medical device or the comparator.

NOTE 2: This definition includes events related to the procedures involved.

NOTE 3: For users or other persons, this definition is restricted to events related to the use of investigational medical devices.

**Anticipated Adverse Events** – Anticipated adverse events are adverse events that have been identified as adverse events related to the investigational device or study procedure. The anticipated events of this clinical investigation are outlined in tDCS Adverse Events Questionnaire (AEQ). The frequency and severity of anticipated AEs will be captured using AEQ.

Anticipated adverse events are:

- Headache
- Neck pain
- Scalp pain
- Tingling
- Itching
- Burning sensation
- Skin redness
- Sleepiness
- Trouble concentrating
- Acute mood change

**Adverse Device Effect (ADE)** – An adverse device effect (ADE) is any adverse event related to the use of an investigational device. This definition includes:

Protocol version: 9



- Adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.
- Any event resulting from use error or from intentional misuse of the investigational medical device.
- "Comparator" if the comparator is a medical device.

# **Serious Adverse Event (SAE)** – A Serious Adverse Event is an AE which:

- 1. Led to a death,
- Led to serious deterioration in the health of the subject, users, or other persons that either resulted in:
  - a) A life-threatening illness or injury, or
  - b) A permanent impairment of a body structure or a body function including chronic diseases, or
  - c) In-patient or prolonged hospitalization, or
  - d) Medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
- 3. Led to fetal distress, fetal death or a congenital abnormality or birth defect including physical or mental impairment (not anticipated in this study as pregnant women are excluded from the study).

NOTE: Planned hospitalization for any pre-existing condition, or a procedure required by the Clinical Investigation Plan, without a serious deterioration in health, is not considered a serious adverse event.

**Serious Adverse Device Effect (SADE)** – a Serious Adverse Device Effect is an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

**Anticipated Serious Adverse Device Effect (ASADE)** – an Anticipated Serious Adverse Effect is an effect which by its nature, incidence, severity, or outcome has been identified in the risk analysis report.

**Unanticipated Serious Adverse Device Effect (USADE)** – this is a serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the current version of the risk analysis report. This is also referred to as an Unanticipated Adverse Device Effect (UADE) in the US. See Section 19.2.4 for details regarding determination and reporting requirements in the US.

**Device Deficiency (DD)** - A device deficiency is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. Device deficiencies include malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling.



Protocol version: 9



**Malfunction** – Failure of an investigational medical device to perform in accordance with its intended purpose when used in accordance with the instructions for use or protocol.

**Use Error** – User action or lack of user action while using the medical device that leads to a different result than that intended by the manufacturer or expected by the user.

NOTE1: Use error includes the inability of the user to complete a task.

NOTE 2: Use errors can result from a mismatch between the characteristics of the user, user interface, task or use environment.

NOTE 3: Users might be aware or unaware that a use error has occurred.

NOTE 4: An unexpected physiological response of the patient is not by itself considered a use error.

NOTE 5: A malfunction of a medical device that causes an unexpected result is not considered a use error.

19.2 CLASSIFICATION OF AN AE

### 19.2.1 SEVERITY

Investigators will assess the severity of the adverse event and classify it according to the following definitions:

- **Mild**: Awareness of a sign or symptom that does not interfere with the patient's usual activity or is transient, resolved without treatment and with no sequelae.
- Moderate: Interferes with the patient's usual activity and/or requires symptomatic treatment.
- **Severe**: Symptom(s) causing severe discomfort and significant impact on the patient's usual activity and requires treatment.

These definitions are for descriptive purposes only and are independent of the judgment of whether an event is classified as an AE or an SAE.

19.2.2 Assessment of Relationship to Use of the Investigational Device or Procedure

The relationship between the use of the medical device (including the medical - surgical procedure) or control procedure the occurrence of each unanticipated adverse event shall be assessed and categorized. During causality assessment, clinical judgment shall be used, and the Clinical Protocol shall be consulted, as all the foreseeable adverse events and the potential risks are listed and assessed there. The presence of confounding factors, such as concomitant medication/treatment, the natural history of the underlying disease, other concurrent illness or risk factors shall also be considered.

19.2.3 SAE RELATIONSHIP ASSESSMENT

Per MDCG 2020-10/1 (May 2020), Investigators will assess the potential relationship of the SAE to the use of the investigational device (including the surgical procedure) or control procedure and classify the causality of the event according to the following definitions.

Protocol version: 9



- Not Related: Relationship to the device or procedures can be excluded when:
  - the event has no temporal relationship with the use of the investigational device, or the procedures related to application of the investigational device;
  - the serious event does not follow a known response pattern to the medical device (if the response pattern is previously known) and is biologically implausible;
  - the discontinuation of medical device application or the reduction of the level of activation/exposure - when clinically feasible - and reintroduction of its use (or increase of the level of activation/exposure), do not impact on the serious adverse event;
  - the event involves a body-site or an organ that cannot be affected by the device or procedure;
  - the serious event can be attributed to another cause (e.g., an underlying or concurrent illness/ clinical condition, an effect of another device, drug, treatment, or other risk factors);
  - the event does not depend on a false result given by the investigational device used for diagnosis, when applicable;
  - harms to the subject are not clearly due to use error;
  - In order to establish the non-relatedness, not all the criteria listed above might be met at the same time, depending on the type of device/procedures and the serious adverse event.
- Possible: The relationship with the use of the investigational device or the relationship with
  the procedure is weak but cannot be ruled out completely. Alternative causes are also
  possible (e.g., an underlying or concurrent illness/ clinical condition or/and an effect of
  another device, drug, or treatment). Cases where relatedness cannot be assessed or no
  information has been obtained should also be classified as possible.
- Probable: The relationship with the use of the investigational device or the relationship with the procedure, seems relevant and/or the event cannot reasonably be explained by another cause.
- Causal Relationship: The serious adverse event is associated with the investigational device or with procedures beyond reasonable doubt when:
  - the event is a known side effect of the product category the device belongs to or of similar devices and procedures;
  - the event has a temporal relationship with investigational device use/application or procedures;
  - the event involves a body-site or organ that
    - the investigational device or procedures are applied to;
    - the investigational device or procedures have an effect on;
  - the serious event follows a known response pattern to the medical device (if the response pattern is previously known);



Protocol version: 9



- the discontinuation of medical device application (or reduction of the level of activation/exposure) and reintroduction of its use (or increase of the level of activation/exposure), impact on the serious event (when clinically feasible);
- other possible causes (e.g., an underlying or concurrent illness/ clinical condition or/and an effect of another device, drug, or treatment) have been adequately ruled out;
- harm to the subject is due to error in use;
- the event depends on a false result given by the investigational device used for diagnosis, when applicable;
- In order to establish the relatedness, not all the criteria listed above might be met at the same time, depending on the type of device/procedures and the serious event.

Where the Investigator or Sponsor remains uncertain about classifying the event, it should not exclude the relatedness and the Investigator should classify the event as "Possibly Related".

### 19.2.4 SAE REPORTING

Flow Neuroscience AB is responsible for the classification and reporting of adverse events and ongoing safety evaluation of the clinical investigation in line with ISO 14155:2020 and US/UK regulatory requirements.

Investigator will report "to the Sponsor, without unjustified delay, all serious adverse events and device deficiencies that could have led to a serious adverse device effect; this information shall be promptly followed by detailed written reports" [ISO 14155:2020 § 9.8 b]. Device malfunctions and use errors should also be reported without unjustified delay.

In the event of becoming aware of any SAE (including all device deficiencies), anticipated or unanticipated, the Investigator will report the event to Flow Neuroscience AB and Curebase immediately (at least within 24 hours after first knowledge of the event) by entering SAE information in the EDC. In the event the EDC is unavailable for any reason, notification to Flow Neuroscience AB should be made via email as follows:

Sponsor Contact: Erik Rehn

E-mail: erik@flowneuroscience.com

Phone: +46736607170

The Investigator should provide additional information on the SAE by updating the information in the EDC as updates become available. Flow Neuroscience AB may also ask for additional clinical reports including redacted source documents to be provided by the Investigator to assist in the assessment of the event. Significant new information and updates should continue to be submitted promptly to and entered in the EDC as they become available, and the Investigator should follow the SAE until it is resolved, or no further improvement is expected.

It is the responsibility of each Investigator to report all SAEs and/or SADEs to the IRB/EC, according to national regulations and IRB/EC requirements. A copy of the IRB/EC report should be



Protocol version: 9



forwarded to Flow Neuroscience AB. In countries that require the Sponsor to report safety events rather than investigators, the Sponsor (Flow Neuroscience AB) will report SAEs and/or SADEs to the EC.

Flow Neuroscience AB will ensure that all SAEs and device deficiencies that could have led to a SAE are reported to the Competent Authorities in accordance with European Medical Devices directives and all applicable national regulations.

Flow Neuroscience AB will ensure that all events that meet the vigilance requirements as described in MDCG 2020-10/1 (Safety reporting in clinical investigations of medical devices under the Regulation (EU) 2017/745) are reported to the Competent Authorities in accordance with European Medical Devices directives and all applicable national regulations.

19.2.5 DETERMINATION AND REPORTING OF UNANTICIPATED ADVERSE DEVICE EFFECTS (US SITES)

The Sponsor shall review all reported SAEs to evaluate whether they meet the criteria for an Unanticipated Adverse Device Effect. For adverse events that are determined to be UADEs, the Sponsor will submit an expedited safety report to the FDA's Center for Devices and Radiological Health (CDRH). The expedited safety report will be submitted to the FDA as soon as possible and, in no event, later than ten (10) business days after the Sponsor first receives notice of the UADE. A copy of this safety report will be provided to all participating study Investigators.

If, following receipt and investigation of follow-up information regarding an adverse event that was previously determined not to be a UADE, the Sponsor determines that the event does meet the requirements for expedited reporting, the Sponsor will submit a report as soon as possible, but in no event later than **ten (10) business days** after this is determined.

19.3 TREATMENT OF AES

The Investigator will treat all participants who experience an adverse event directly related to the device.

19.4 SAFETY OVERSIGHT: CLINICAL EVENTS COMMITTEE (CEC)

The Clinical Events Committee (CEC) will adjudicate all AEs and protocol deviations. SAEs and AEs deemed "definitely," "probably," and "possibly related" or with an "unknown relationship" to the device or procedure, primary endpoint failure, and the following neurological AEs, including neurologic deterioration will be reviewed.

19.5 SAFETY/SUICIDE RISK MANAGEMENT PLAN

All study participants will be provided a safety crisis action plan for suicide risk at the time of study enrollment. The crisis action plan will include the following information;

- Name, address, and telephone number of the closest hospital emergency department near the study participant's residence
- Contact details of next of kin/friends for support
- Study participant's regular treating physician's name and contact information



- National Suicide Prevention Lifeline 800-273-8255
- Strategies for coping with suicidal ideation/crisis.
- Further, subjects will be notified that study personnel will contact their psychiatrist in the case of worsening depression/suicidality (worsening depression is defined as 30% increase in HDRS-17 score compared to baseline).

All participants will be informed about the warning signs of suicidal ideation and behavior at the start of the study. Throughout the study, subjects will be monitored by study psychiatrists.

If the C-SSRS questions 4, 5, and 6b are positive during the study assessments, the participant will be asked to go to the nearest emergency department or mental health crisis center.

The suicide risk management plan document (attachment "Brown\_StanleySafetyPlan") will be completed with patients.

### 20 STOPPING RULES

The following events will result in the study stopping:

- If two subjects commit suicide
- If three subjects attempt suicide
- If ≥ 2 serious adverse events (SAEs) occur that are device-related, as determined by investigators, the IRB, the FDA, or the Clinical Events Committee (CEC)

If any of the stopping rules are reached, enrollment will be paused and the FDA will be notified in a supplement to enable review of the information.

#### 21 CLINICAL MONITORING

#### 21.1 SITE MONITORING

The study will be monitored to ensure that it is conducted in conformance with the monitoring plan by an independent CRO to assess continued compliance with the protocol, recognized Good Clinical Practices, FDA's 2013 guidance document "Guidance for Industry Oversight of Clinical Investigations — A Risk-Based Approach to Monitorings, and federal regulations outlined in 21 CFR Part 812

- Subpart A
- Subpart B
- Subpart C -
  - 812.3 Definitions
  - 812.25 Investigational Plan
  - 812.28 Acceptance of data from clinical investigations conducted outside the United States

T1 Effective Date: 19FEB2021

Protocol version: 9

- 812.30 FDA action on applications
- 812.35 Supplemental applications
- 812.36 Treatment use of an investigational device



Protocol version: 9



- 812.40 General responsibilities of sponsors
- 812.43 Selecting investigators and monitors
- 812.46 Monitoring investigations
- 812.47 Emergency research under 50.24 of this chapter
- 812.140 Records
- 812.150 Reports

In addition, the monitor verifies that study records are adequately maintained, that data are reported in a satisfactory manner with respect to timeliness, adequacy, and accuracy, and that the Investigator continues to have sufficient staff and facilities to conduct the study safely and effectively.

The study may also be subject to a quality assurance audit by the Sponsor or its designees, as well as inspection by appropriate regulatory authorities. It is important that the Investigator and relevant study personnel are available during on-site monitoring visits or audits and that sufficient time is devoted to the process.

The organization responsible for monitoring the study is:

Curebase Inc. 335 S Van Ness Ave San Francisco, CA 94103-3627 (519)590-8490 www.curebase.com

In addition to ensuring adequate communication between the Investigators and the Sponsor, the CRO's duties include on-site visits and review of study documents and reported data. The CRO study representatives will be provided with appropriate device and protocol training prior to the study and will follow a Monitoring Plan for all study-related monitoring activities.

## 21.2 Monitoring Activities

Monitoring visits include a pre-study Site Initiation Visit, periodic Interim Monitoring Visits, and a Close-Out Visit at the end of the site's participation in the study.

Each site's Investigator will allocate adequate time for monitoring activities. The Investigator will also ensure that the monitor or other compliance or quality assurance reviewer is given access to the study-related documents and study-related facilities and has adequate space to conduct the monitoring visit.

Monitoring visits will be documented on monitoring visit reports, and will aim to verify that:

- Compliance with the clinical protocol and applicable regulations is being maintained
- Source data is verified and signed-off upon as accurate



Protocol version: 9



- Participant files are accurate and complete
- Participant withdrawal has been documented (if applicable)
- Participant non-compliance has been documented (if applicable)
- The Investigator and site staff are informed and knowledgeable of all relevant document updates concerning the clinical investigation
- Only authorized individuals are performing study-related functions
- The investigational device is being used according to the protocol and instructions for use
- Adequacy of staffing and facilities
- Signed and dated ICFs have been obtained from each participant
- eCRFs and queries are complete
- All adverse events are reported to the Sponsor
- All serious and unanticipated adverse device events are reported to the Sponsor and the IRB/EC
- All other required IRB/EC reports, notifications, applications, submissions, and correspondence are maintained in the Investigator's files and are accurate
- Corrective and preventive actions have been implemented (if applicable)

## 21.3 Frequency of Visits

To ensure that the study is conducted in accordance with the terms of the clinical protocol, study monitors must visit each investigational site at routine intervals throughout the duration of the study. The exact frequency of visits shall be determined on an individual site basis as detailed in the Clinical Monitoring Plan, and shall depend upon the following factors:

- Rate of participant enrollment
- Experience of the Investigator in conducting clinical studies
- Record of previous site compliance

# 21.4 AUDIT AND INSPECTIONS

Participation as an Investigator in this study implies acceptance of potential inspection by government regulatory authorities. The Investigator must also be prepared to permit study-related audits and inspections by the Sponsor, CRO, IRB/EC and the site's institutional compliance and quality assurance groups. The Investigator will ensure the capability for inspections of applicable study-related facilities, records, and reports.

Protocol version: 9



# 22 STATISTICAL ANALYSIS

# 22.1 STUDY HYPOTHESIS

The primary clinical outcome of the study will be to compare the adjusted mean group differencebased on HDRS-17 scores of the two arms at 10 weeks compared to baseline.

The primary efficacy hypothesis is the change in HDRS-17 scores between 10 weeks and baseline between subjects randomized to the study device relative to those subjects randomized to Sham. The formal statistical hypothesis is as follows:

Ho:  $d_{flow} - d_{sham} \le 0$ Ha:  $d_{flow} - d_{sham} > 0$ 

Where  $d_{flow}$  and  $d_{sham}$  are the adjusted mean group difference in HDRS-17 scores in subjects randomized to Flow and Sham groups, respectively.

# 22.2 SAMPLE SIZE ASSUMPTIONS AND CALCULATIONS

The sample size calculation is based on data from Brunoni et al (2017). The calculation is based on a two- sample t-test for mean difference with the following assumptions:

- Group difference in means = 3.2
- Standard deviation of Investigational and Sham groups = 7.1 and 7.9, respectively
- One-sided type I error = 0.025
- 80% power

The resulting sample size is 176 subjects. To obtain an increase in statistical power (87.6%), 216 subjects were chosen. Accounting for 20% attrition, the overall sample size will be 270 subjects.

# 22.3 STUDY POPULATIONS

# 22.3.1 INTENT-TO-TREAT ANALYSIS SET (ITT)

All randomized subjects will be included in the "intent-to-treat" (ITT) analysis set and classified according to their intended treatment regardless of failure to complete the required follow-up examinations. Subjects excluded prior to randomization will be considered screening failures.

## 22.3.2 As Treated Analysis Set (AT)

The As Treated Analysis Set (AT) will consist of ITT subjects who receive at least 1 treatment of study device (Active or Sham). Subjects will be analyzed according to the study treatment received. The As Treated Analysis Set will be used for all summaries of safety and tolerability data.

## 22.3.3 Modified Intent-to-Treat Analysis Set (MITT)

The modified intent-to-treat (mITT) analysis set will include ITT subjects who receive at least 1 treatment of study device (Active or Sham) and will exclude patients who were randomized in error. The number of exclusions from the mITT analysis set is expected to be small and will only be

Protocol version: 9



based on information that was known or could have been known prior to the first treatment. Subjects in the mITT population will be analyzed in the group to which they were randomized.

22.3.4 PER PROTOCOL ANALYSIS SET (PP)

The Per Protocol (PP) analysis set will be comprised of the following:

- Subjects in the mITT analysis set
- Subjects with device failure within the 10-week follow-up period
- Subjects with deviation from the clinical investigation plan is caused by the investigational device or by problems with respect to tolerability

Subjects who will be excluded from the PP analysis set are as follows:

- Subjects with major protocol violations that would be expected to confound clinical assessment during follow-up as determined by the PIs.
- Subjects who took new pharmaceutical substances or treatments during the clinical investigation which are listed as an exclusion criteria;
- Subjects who do not meet the inclusion criteria or exclusion criteria.
- Users who have performed less than 10 sessions (300 minutes) during the first 3 weeks will be excluded from the analysis.

Subjects in the PP population will be analyzed in the group to which they were randomized.

# 22.4 RANDOMIZATION

After a subject has met all inclusion criteria and none of the exclusion criteria, and creates an account in the Flow app, the subject will be randomized. Randomization will be performed in a 1:1 ratio to the Active and Sham groups. Randomization will be performed using randomly permuted block sizes of 4 and 6 and done independently for the two sites.

## 22.5 Testing of Primary Effectiveness Hypotheses

The primary effectiveness endpoint is the change in adjusted mean group difference in the HDRS-17 scores between 10 weeks and baseline between subjects randomized to the active study device relative to those subjects randomized to sham. The formal statistical hypothesis is as follows:

$$H_o$$
:  $d_{flow} - d_{sham} \le 0$   
 $H_a$ :  $d_{flow} - d_{sham} > 0$ 

Where  $d_{\text{flow}}$  and  $d_{\text{sham}}$  are the adjusted mean group difference in HDRS-17 scores in subjects randomized to Active and Sham groups, respectively.

The mITT population will be the analysis population used to analyze the primary effectiveness endpoint. The endpoint will be analyzed when all randomized subjects have completed their 10-week visit, been withdrawn



Protocol version: 9



from the trial or passed the end of their 10-week follow-up visit window. The difference in the group mean differences will be assessed using a mixed model for repeated measures. If the p-value of the difference in the group mean differences is less than one-sided p= 0.025, then the trial declared a success.

#### 22.5.1 Multiple Imputation Analysis

The mixed model for repeated measures (MMRM) allows for inclusion of patients with missing Week 10 values. If all subjects have at least one follow-up evaluation, the following MMRM will be utilized for the primary superiority test. If there are subjects without at least one post baseline assessment, the multiple imputation analysis summarized below will be the primary analysis method. Least squares estimated values from the MMRM will be reported for HDRS-17 at each visit and as such these estimates include implicit imputations of missing values.

Details of the MMRM used to evaluate the primary endpoint are described in the attached Statistical analysis plan.

#### 22.6 Missing Data/Sensitivity Analysis

Details of the handling are in the attached Statistical analysis plan.

#### 22.7 Covariates/Covariate Analysis

The heterogeneity of treatment effects for the primary effectiveness endpoint will be examined for subgroups using baseline variables. These will include, but are not limited to, age (split at median), and sex at birth. Subjects on antidepressants and/or psychotherapy drugs during the course of the trial will constitute their own subgroup and be characterized and described in the clinical study report. The mixed model for repeated measures will be run to see the impact of the treatment effect by each subgroup of interest separately. The results will be reported as mean differences and 95% confidence intervals for each subgroup. These results will be graphically displayed in a forest plot.

## 22.8 Secondary Effectiveness Endpoints

Secondary effectiveness endpoints will be analyzed descriptively.

For continuous variables (CONT), results will be summarized with the numbers of observations, means, standard deviation, median, minimums and maximums. Differences between the two groups, where specified, will be summarized with the differences of the two means, and 95% confidence intervals for the difference between the means. These calculations will be done under the assumption that data for the two groups are independent and approximately normally distributed. The confidence interval for the difference of two means will be calculated under the assumption of unequal variances. If the asymptotic assumptions fail, then nonparametric summary statistics (medians, 25th and 75th percentile) may be displayed as an alternative.

For binary variables (BIN), results will be summarized with patient counts, percentages/rates. Differences between the two groups, where specified, will be summarized with the difference in percent and the Newcombe score 95% confidence interval for the difference of two percentages.

For correlation analysis, Spearman correlation will be used to assess the association between two continuous variables. The correlation coefficient and the 95% confidence intervals will be reported.



Protocol version: 9



There are three secondary endpoints controlled multiplicity (see below):

- The mean change in points for MADRS score from baseline to Week 10. This will be evaluated using the same statistical methodology as the primary endpoint.
- Clinical Response will be analyzed as a responder endpoint. Clinical Response is defined as a >50% reduction from the baseline HDRS-17 or MADRS score, MADRS-s at Week 10.
- Remission will be analyzed as a responder endpoint where remission is defined as an HDRS-17 score ≤7 or a MADRS score ≤10). The endpoint will be tested using a two-group large-sample normal approximation test of proportions with a one-sided 0.025 considered significant.
- Quality of life improvement as measured by EQ-5D-3L in the active compared to sham arm at week 10 compared to baseline.

#### 22.9 EXPLORATORY ENDPOINTS

The following list of secondary endpoints will be analyzed using the mITT population and will be summarized based on the type of data: Continuous (CONT), Binary (BIN) or Correlation (CORR):

- Montgomery–Åsberg Depression Rating Scale (MADRS) response rate at all follow-up time points (CONT)
- Montgomery–Åsberg Depression Rating Scale Self-report (MADRS-s) scores of the two arms (response and remission rates) at all time points (CONT)
- Hamilton Anxiety Rating Scale (HAM-A) at all time points (CONT)
- Young Mania Rating Scale (YMRS) at all time points (CONT)
- tDCS Adverse Events Questionnaire (AEQ) at 10 and 20 weeks (CONT)
- HDRS-17 (CONT), MADRS (CONT), MADRS-s mean decrease (CONT), remission (BIN), and response rate (BIN) at 6 weeks comparison between groups.
- HDRS-17 (CONT), MADRS (CONT), MADRS-s (CONT) at 20 weeks (after open-label)
- Correlation between MADRS and MADRS-s. (CORR)
- Correlation between the percent of sessions using the FLOW FL-100 and HDRS-17/MADRS decrease in the active group at 10 weeks.
- The within-patient clinically meaningful improvement as defined as at least -3 points on the HDRS-17 scale. The percentage of subjects for each arm that reaches -3 points or more improvement and also the Cumulative Distribution Function Curves of Change in HDRS-17 Score from Baseline to Primary end-point by arm.

### 22.10 MULTIPLICITY ADJUSTMENT

The secondary endpoints will only be tested if the primary endpoint demonstrates superiority. By pre-specifying the order in which the primary and conditional effectiveness hypotheses are performed, there is no type 1 error inflation and nominal alpha levels may be used on the primary endpoint.

Should the primary endpoint be met, the clinical response endpoint (Endpoint #1 in SAP version 2) will be tested. Should the secondary Endpoint #1 be met, the remaining endpoints will be tested using Hochberg correction for multiplicity. Complete details for multiplicity adjustment are provided in the SAP.

Protocol version: 9



#### 22.11 EVALUATION OF BLINDING

An evaluation of blinding will be performed. Prior to subjects unblinding through the system they will respond to the question "Which treatment arm do you think you are in?" (answers: sham/active), followed by the question "How certain are you of this?", with the options 1 to 5 where 5 is very certain and 1 is very uncertain. The counts and percentages of the subjects responding correctly will be tabulated and reported.

#### 22.12 DEVICE SURVIVAL

Kaplan-Meier survival analysis will be used to characterize device failure time. Device failure in this study is defined as the device not operating as intended without unexpected failure. Unexpected failure is defined as a failure that is not related to device functionality. For example, the device accidentally falling out of a window would be categorized as an unexpected device failure. In contrast, the device failing to turn on would be considered an expected device failure. As the device is not expected to have any unexpected failures, unexpected failures will only be reported if they occur. Lifetables will be tabulated indicating the number of "failures" and the number of "at- risk" subjects over time for all failures, unexpected failures and expected failures. If there are more than one of each expected and unexpected failures, a log-rank test will be performed to compare the device failure time distribution.

#### 22.13 Poolability Analysis

Poolability will be assessed through stratification of the primary endpoint by Country (OUS and US). Within country point estimates will be calculated along with nominal descriptive 95% Confidence Intervals. The focus of this analysis will be on the similarity of the country specific point estimates. Differences will be described in the Clinical Study Report.

Statistical evaluation of the primary endpoint will be evaluated by adding site by treatment group term to the primary MMRM model. A p-value of <= 0.10 will be considered significant for this poolability assessment. Should a significant site x treatment group interaction be present, the patient factors of age, gender, and baseline scores will be assessed to understand if differences in case-mix factors explain differences observed between sites.

#### 22.14 SAFETY ANALYSES

Assessment of the safety of the investigational device will include an evaluation of the incidence and severity of complications and adverse reactions associated with the treatment.

Adverse event rates will be summarized by type of AE and for specific AEs in two ways:

- 1. per subject incidence of specific AEs and classes of AEs and
- 2. by event, summarizing event counts by visit interval over time and in accordance with FDA Guidance (CDRH 2004)<sup>15</sup>.

Device and procedure-related events will be summarized by severity and relatedness. Events listings that include details such as relatedness, severity, onset, and resolution status will be provided for all events and relevant subsets of events such as serious events and related events. Primary safety comparisons will be performed using the AT analysis set. The summary tables will show the adverse events (in coded terms), the total number of events, and the number and the percentage of subjects affected in each treatment group

<sup>&</sup>lt;sup>15</sup> CDRH. Guidance for Industry and FDA Staff: Clinical Data Presentations for Orthopedic Device Applications, December 2, 2004.



Protocol version: 9



("subject wise evaluation") and stratified by relation to device and severity. Data of dropouts will be presented separately, and possible bias will be discussed in the final report.

All AEs will be summarized in listings for the AT analysis set. The following AE listings will be constructed:

- AE Listing 1 All AEs Sorted by Group and Event Type
- AE Listing 2 All AEs Sorted by Group and Subject
- AE Listing 3 Serious AEs
- AE Listing 4 Severe AEs
- AE Listing 5 Device Related AEs
- AE Listing 6 Serious Device Related AEs
- AE Listing 7 Severe Device Related AEs
- AE Listing 8 Other AEs
- AE Listing 9 AEs among subjects discontinued early
- AE Listing 10 AEs among subjects who died

## 22.15 INTERIM ANALYSES

An interim analysis testing for futility, sample size re-estimation, and claiming study success with a sample size smaller than the maximum specified is specified. Please see the details in the Adaptive Design Report detailing all elements of this process.

## 23 Ethics & Protection of Human Subjects

#### 23.1 ETHICAL REVIEW

The study will be performed in accordance with the standard guidance on clinical investigations with medical devices on human subjects and recommendations guiding physicians in biomedical research involving human subjects adopted by the 18th World Medical Assembly, Helsinki, Finland, 1964 and later revisions.

The clinical investigational plan, informed consent, any other study specific study documents as required by regulations and all amendments to these study documents will be reviewed and approved by the FDA and appropriate IRB/EC before enrollment of any patient. In addition, the sponsor will keep the regulatory authorities informed of any SAEs throughout the study course, if applicable.

#### 23.2 REGULATORY CONSIDERATIONS

This study will be conducted in accordance with the Good Clinical Practice (GCP) guidelines and other applicable regulatory requirements including but not limited to:

- FDA Regulations on Investigational Device Exemption (21 CFR 812)
- FDA Regulations on research with human beings (21 CFR 50, 54 and 56)
- Health and Human Services (DHHS) Regulations on research with human beings (45 CFR 46 Subparts A, B, C, and D)



Protocol version: 9



- International Conference on Harmonization (ICH) Guidance for Industry-E6 Good Clinical Practice: Consolidated Guideline
- The Declaration of Helsinki

## 23.3 STUDY AMENDMENTS

All changes to the protocol that impact validity of data, scientific soundness, the rights safety, or welfare of the participants, must be documented in the format of an amendment with justification statements in the cover letter to the IRB/EC and FDA. All amendments must be submitted to the IRB/EC and regulatory authority for review and approval. Following approval, the protocol amendment will be distributed to all protocol recipients at each investigational site.

## 23.4 INSURANCE

The Sponsor has issued clinical trial insurance with appropriate coverage for the continuation of the entire study.

#### 24 Data Handling and Recordkeeping

### 24.1 EDC AND ECRFs

eCRFs will be completed in a 21 CFR Part 11 compliant electronic data capture (EDC) system for each patient enrolled into the clinical study. The study coordinator will enter the source data onto the eCRFs, and study monitors will verify that the source documents match the eCRFs. Once verified, the study monitor will lock the field via a monitoring approval step so the data cannot be changed unless requested.

All procedures for the handling and analysis of data will be conducted using good clinical data management practices within systems meeting FDA guidelines for the handling, storage, and analysis of data for clinical studies.

The Investigator will sign off on the Eligibility Criteria, all Adverse Event, Protocol Deviation and Study Completion eCRFs and will sign each patient's casebook once the patient completes the study to attest that all data entered on the eCRFs are complete and accurate. All of the above signatures will be completed digitally within the EDC system using the system's Part 11 compliant digital signature system function.

Any required data clarifications will be handled within the EDC system's query management system. The EDC will be programmed to automatically place data clarification queries on missing values and values out of acceptable ranges. Study monitors and data managers will also be able to add data clarification queries to data points within the system. Study coordinators will have the opportunity to correct data and/or respond to the query for review by monitors and data managers.

Protocol version: 9



# 24.2 CAPTURE OF PATIENT REPORTED OUTCOMES

Patient reported outcomes (PROs) will be collected via the participant's personal smartphone or other device running Android 5.0+ or iOS 12+ and the data will be transmitted directly into the EDC. As the data is originated in the participant's device, it is considered to be electronic source and the data is automatically locked as soon as it enters the EDC to ensure that it is secure.

## 24.3 Study Records Retention

The Investigator and the Sponsor will maintain accurate, complete, and current records relating to participation in this clinical investigation. If the Investigator wishes to assign the responsibility of maintaining the study files to someone else or move them to another location, he/she should consult with the study sponsor in writing regarding the change. The Investigator will take measures to ensure that these essential documents are not accidentally damaged or destroyed.

Upon study completion, the study files must be maintained in a known location for a maximum of a 2 years following the date a marketing application is approved for the medical device for the indication for which it is being investigated; or, if no application is to be filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and FDA is notified.

The Investigator and Sponsor will maintain records in accordance with 21 CFR 812, Subpart G, to include:

- Current and past versions of the IRB/EC-approved clinical protocol and amendments and corresponding IRB/EC-approved consent form(s) and, if applicable, participant recruitment advertisements
- FDA correspondence related to the IDE application; including supplemental IDE applications, current investigator lists, progress reports
- IRB/EC correspondence (including submissions and approval notifications) including safety and protocol deviation reports, and annual or interim reports
- Signed Clinical Trial Agreement
- Signed Investigator Agreements and financial disclosure forms for participating Investigators
- Curriculum vitae (Investigator and Sub-Investigators)
- Certificates of required training for Investigators and Sub-Investigators, including human subject protection and Good Clinical Practice
- Instructions for handling the investigational device and other study-related materials
- Device tracking logs
- Signed ICFs



Protocol version: 9



- eCRF and Source Documents
- Monitoring visit confirmation and follow-up letters
- Copies of relevant Sponsor-Investigator correspondence, including notifications of adverse event information
- Screening and Enrollment Log
- Signed informed consent forms
- Final clinical study report

#### 24.4 Publication and Data Sharing Policy

Data generated from the conduct of this study will be used to support an application by Flow Neuroscience AB as an original Premarket Approval (PMA) from FDA. Publication of the results of the study will follow Flow Neuroscience AB 's Publication and Presentation Policy.

# 24.5 PARTICIPANT AND DATA CONFIDENTIALITY

Participant confidentiality will be maintained throughout the study in a way that ensures that data can always be tracked back to the source data. For this purpose, a unique participant identification code (two-digit site identification number and three-digit participant name identification number code assigned sequentially) will be used that allows identification of all data reported for each participant without traceability back to the actual participant.

The Principal Investigator or institution shall provide direct access to source data during and after the clinical investigation for monitoring, auditing, IRB/EC review and regulatory authority inspections.

For investigational sites within the United States, "Protected Health Information" will be treated and maintained in compliance with the Health Insurance Portability and Accountability Act of 1996 (HIPAA) Privacy rule.

The duration of storage time of personal data at the investigational sites will be in accordance with national regulations. Electronic Case Report Form (eCRF) data captured and maintained in Curebase for each participant. Curebase stores all data in a secure cloud server of Amazon Web Services (AWS) and complies with most of HIPAA and GDPR standards, including but not limited to: password protection, platform encryption, and 2-factor verification. Curebase takes as much action as possible to maximize the protection and security of subjects' sensitive information. All data pertaining to a clinical study, including protected health information (PHI), will be retained for the duration of the study, and for 2 years thereafter, in compliance with FDA monitoring obligations. At this point, the identifiable PHI obtained during the study will be deleted. Curebase will share pseudonymized data collected from subjects with authorized representatives.

After 2 years have elapsed since the completion of a clinical investigation, Curebase will retain a de-identified version of the data obtained during that study. Curebase may retain this data

Protocol version: 9



indefinitely and may use it for a variety of purposes that will include, but not be limited to, making improvements to the Curebase product.

Information obtained while executing this study, including still and motion photography, may be presented for regulatory, clinical, or educational purposes if no participant is identified. The data collected is the property of Flow Neuroscience AB.

## 24.6 Investigator Records

The investigator is responsible for the preparation and retention of the records cited below. All these records, except for participant's case history records, should be filed in the Investigator Site File.

#### 24.7 Participant Records

- All Source Documentation Worksheets
- Supporting data (e.g., medical records, clinic charts)

## 24.8 INVESTIGATOR RECORDS AND REPORTS

The investigator is responsible for the timely preparation and submission of the reports cited below.

Table 5: Investigator Reports

| Report | Sent To | Timing of Report |
|---|---|---|
| Unanticipated | Flow | UADE must be reported as soon as possible, but in no |
| adverse device | Neuroscience | event later than 10 business days after the investigator |
| effect (UADE) | AB, IRB/EC | first learns of the event |
| Withdrawal of | Flow | Reported within 5 business days |
| IRB/EC | Neuroscience | |
| approval | AB | |
| Progress | Flow | Reported as requested by Flow Neuroscience AB or the |
| reports | Neuroscience | reviewing IRB/EC, but at least yearly |
| | AB, IRB/EC | |
| Deviations<br>from the<br>investigation<br>plan | Flow<br>Neuroscience<br>AB, IRB/EC<br>(FDA) | A deviation to protect the life or physical well-being of a participant in an emergency must be reported no later than 5 business days after the emergency occurred. Deviations that may affect the scientific soundness of the investigational plan or the rights, safety, or welfare of the participant (and are not an emergency) must receive prior approval by Flow Neuroscience AB and be reported to the FDA and IRB/ECs. |
| Device use without informed consent | Flow<br>Neuroscience<br>AB, IRB/EC | This deviation must be reported within 5 business days after the use occurs. |



Protocol version: 9



| Final Report | Flow | This report must be submitted within 3 months after |
|---|---|---|
| | Neuroscience | termination or completion of the investigation or the |
| | AB, IRB/EC | investigator's part of the investigation. |
| Other | FDA, IRB/EC | Upon request, accurate, complete, and current |
| | | information about any aspect of the investigation must be |
| | | reported. |